# ADDENDUM STATISTICAL ANALYSIS PLAN

(Protocol No. ASN100-201)

A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety and Efficacy of a Single Dose of ASN100 for the Prevention of *Staphylococcus aureus* Pneumonia in Heavily Colonized, Mechanically Ventilated Subjects

#### **DEVELOPMENT PHASE: 2**

#### **Sponsor:**

Arsanis, Inc. 890 Winter Street, Suite 230 Waltham, MA 02451-1472

**SAP Addendum Version:** 1.0

**Date:** October 25, 2018

#### CONFIDENTIAL

This material is the proprietary property of Arsanis, Inc. The information is confidential and is to be used only in connection with matters authorized by Arsanis, Inc. No unpublished information presented in this document is to be disclosed to others without prior written permission from Arsanis, Inc.

## Statistical Analysis Plan Approval:

This Statistical Analysis Plan has been reviewed and approved by:

Mei Chen, PhD

Director, Biostatistics

Medpace, Inc.

19 01

Date

Brian S. Murphy, MD MPH FIDSA

Vice-President, Infections Disease

Medpace, Inc.

2500 2018

Date

Chris Stevens, MD

Chief Medical Officer

Arsanis, Inc.

10/25/201 Date

Date

Ed Campanaro

Senior Vice President, Clinical Operations

Arsanis, Inc.

Date

# TABLE OF CONTENTS

| TABLE | OF CONTENTS | 3 |
|--------|----------------------------------------------|----|
| 1. | LIST OF ABBREVIATIONS | 4 |
| 2. | INTRODUCTION | 6 |
| 3. | STUDY METHODS | 7 |
| 3.1. | Analysis Populations | 7 |
| 3.1.1. | Intent-to-Treat Population (ITT) | 7 |
| 3.1.2. | Modified Intent-to-Treat Population (MITT) | 7 |
| 3.1.3. | Per Protocol (PP) Population | 7 |
| 3.1.4. | Safety Population | 8 |
| 3.2. | Subject Disposition | 8 |
| 3.3. | Demographic and Baseline Characteristics | 8 |
| 3.4. | Prior and Concomitant Medications/Procedures | 9 |
| 3.5. | Analysis of Efficacy | 9 |
| 3.5.1. | Primary Efficacy Endpoint | 9 |
| 3.5.2. | Additional Analyses for S. aureus Pneumonia | 10 |
| 3.5.3. | Secondary Efficacy Endpoints | 11 |
| 3.5.4. | Exploratory Efficacy Endpoints | 11 |
| 3.6. | Subgroup Analyses | 12 |
| 3.7. | Analysis of Safety Data | 13 |
| 3.7.1. | Adverse Events | 13 |
| 3.7.2. | Vital Signs | 14 |
| 3.7.3. | Clinical Laboratory Tests | 14 |
| 4. | GENERAL INFORMATION | 15 |
| 4.1. | Statistical Software | 15 |
| 4.2. | Format of Tables, Listings, and Figures | 15 |
| 5. | APPENDIX | 16 |

## 1. LIST OF ABBREVIATIONS

| AE | Adverse event |
|---|---|
| ALT | Alanine aminotransferase |
| ALP | Alkaline phosphatase |
| ASN-1 | Broadly cross-reactive anti-toxin monoclonal antibody that targets alpha-hemolysin (Hla) and 3 F-components (HlgB, LukF, LukD) involved in forming 4 of the 5 bi-component leukocidins of <i>Staphylococcus aureus</i> |
| ASN-2 | Anti-toxin monoclonal antibody that targets the fifth bi-component leukocidin of <i>Staphylococcus aureus</i> , LukGH |
| ASN100 | A combination of the 2 fully human monoclonal antibodies ASN-1 and ASN-2 |
| AST | Aspartate aminotransferase |
| ATC | Anatomical therapeutic chemical |
| BMI | Body mass index |
| CSR | Clinical study report |
| ETA | Endotracheal aspirate |
| HABP | Hospital-acquired bacterial pneumonia |
| ICF | Informed consent Form |
| ICU | Intensive care unit |
| ITT | Intent-to-Treat |
| LLN | Lower limit of normal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MITT | Modified Intent-to-Treat |
| POP | Population and outcome plan |
| PP | Per Protocol |
| PT | Preferred term |
| S. aureus | Staphylococcus aureus |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SDO | Sponsor-defined outcome |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| TFLs | Tables, figures, and listings |
| ULN | Upper limit of normal |

25OCTOBER2018 

| VABP | Ventilator-associated bacterial pneumonia |
|------|-------------------------------------------|
| WHO | World Health Organization |

25OCTOBER2018 

## 2. INTRODUCTION

This Addendum to the Statistical Analysis Plan (SAP) describes the final selected analyses and reporting based on the final SAP (dated June 25, 2018, Version 1.0), and as outlined in appendix Section 5, the final tables, figures, and listings (TFLs) shells. The purpose of this Addendum is to outline the subset of analyses to support the completion of the Clinical Study Report (CSR) for Protocol ASN100-201.

25OCTOBER2018 

#### 3. STUDY METHODS

### 3.1. Analysis Populations

The following analysis populations will be used for analyses.

#### **3.1.1.** Intent-to-Treat Population (ITT)

The ITT Population includes all subjects who are randomized to receive study drug.

#### **3.1.2.** Modified Intent-to-Treat Population (MITT)

The MITT Population includes all subjects in the ITT Population who receive study drug and who are heavily colonized with *S. aureus* as determined by quantitative or semi-quantitative culture of an ETA specimen. Exclusion from the MITT Population will be determined programmatically for each ITT subject. Programmatically determined assignment into the MITT Population will be evaluated for confirmation or Sponsor Override as applicable during a Review Meeting of the Population and Outcome Plan (POP) Review Group, as described in the POP.

Review Meetings will be held on a regular basis throughout the conduct of the study. The number of subjects included in each Review Meeting will vary depending on the number of subjects included in a data review cycle per the Medpace Rolling Data Lock Plan.

The final MITT Population classification will be performed in a blinded fashion and prior to final database lock and unblinding. After the Review Group's review, any Sponsor overrides of the MITT Population flags will be finalized and documented. The MITT Population flags will be included in the analysis datasets.

#### 3.1.3. Per Protocol (PP) Population

The PP Population includes all subjects in the MITT Population who also meet the following criteria:

- Did not have any major protocol violations that would affect assessment of efficacy based on medical review of available data:
- Randomized in a timely manner following collection of an ETA specimen showing heavy *S. aureus* colonization;
- Was mechanically ventilated at randomization;
- Had an appropriate chest image performed at randomization;
- Did not have a change of oxygenation and onset of purulent secretions at randomization;
- Was not diagnosed with pneumonia at randomization or within 24 hours of receiving study drug;
- Received an adequate dose of study drug administered in a timely manner following study drug preparation,

25OCTOBER2018 

- Did not die within 24 hours of receiving study drug;
- Did not have Investigator Diagnosis of Pneumonia within 24 hours of receiving study drug; and
- Complete an adequate number of Monitoring Period assessments through Day 22 based on medical review of available data.

Exclusion from the PP Population will be determined programmatically for each MITT subject. Programmatically determined assignment into the PP Population will be evaluated for confirmation or Sponsor Override as applicable during a Review Meeting.

The final PP Population classification will be performed in a blinded fashion and prior to final database lock and unblinding. After the Review Group's review, any Sponsor Overrides of the PP Population flags will be finalized and documented. The PP Population flags will be included in the analysis datasets.

#### 3.1.4. Safety Population

The Safety Population includes all subjects who receive any amount of study drug and have at least 1 post-treatment safety assessment.

### 3.2. Subject Disposition

Subject disposition will be summarized for the ITT Population for each treatment group and in total. The following subject disposition categories will be included in the summary for the ITT Population:

- Subjects who randomized in primary prevention study,
- Subjects who randomized in treatment sub-study,
- Subjects who received any study drug,
- Subjects who completed the study assessments through Day 22,
- Subjects who did not complete the study assessments through Day 22,
- Subjects who completed the study assessments through Day 90,
- Subjects who did not complete the study assessments through Day 90, and
- Subjects who completed assessments through Day 22, but did not complete the study assessments through Day 90.

For subjects who did not complete the study assessments through Day 90, a summary will be provided by reason of discontinuation. In addition, the total number of subjects for each defined population will be tabulated.

# 3.3. Demographic and Baseline Characteristics

Demographic information including sex, race, ethnicity, corrected randomization stratification factor (receipt or non-receipt of concomitant anti-staphylococcal antibiotics at the time of randomization that are potentially active against *S. aureus* pneumonia), age

25OCTOBER2018 

(as a continuous variable and categorized as <55, 55 - <65, 65 - <75 and  $\geq$ 75 years, and categorized as <50, 50 - <65, and  $\geq$ 65 years), height, weight, and BMI (as a continuous variable, categorized as <25, 25 - <30, 30 - <35, and  $\geq$ 35 kg/m2), type of hospital unit at time of ICF (ICU and non-ICU), type of ICU, Length of stay (total days) in ICU post-treatment, Length of stay in ICU post-treatment category (<5, 5-12, >12 - 22, and >22 days), Acute kidney injury status at Day 2 visit, baseline creatinine (as a continuous variable and categorized as <2 and  $\geq$ 2 mg/dL), and reason for mechanical ventilation (trauma, cardiovascular impairment, neurological impairment, pulmonary impairment, and other) will be summarized by treatment group for the ITT, MITT, PP, and Safety Populations.

#### 3.4. Prior and Concomitant Medications/Procedures

Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (Sept 2016E B2). Concomitant procedures will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, Version 19.1).

Prior medications are medications used before the initiation of study drug administration. Any medications used on or after the initiation of study drug administration will be included as concomitant medications. Hence medications ongoing at start of study medication will be counted as both prior and concomitant medication.

The number and percentage of subjects taking concomitant medications will be summarized for the ITT Population by anatomic therapeutic chemical (ATC) class and preferred term for each treatment group and overall.

Prior and concomitant medications/procedures will be listed by subject.

# 3.5. Analysis of Efficacy

For all efficacy analyses, subjects will be analyzed in the treatment group to which they were randomized.

Sponsor defined outcomes were determined based on the review of microbiology results from samples tested at the central laboratory. In cases where a sample was not sent to the central laboratory, the determination was based on results from samples tested at the local microbiology laboratory. In all cases where both a local and central result were available, concordance was confirmed in terms of *Staphylococcus aureus*. Therefore, the study analysis utilized local microbiology data in order to utilize a more complete dataset.

#### 3.5.1. Primary Efficacy Endpoint

The primary efficacy endpoint is whether the subject has or has not developed *S. aureus* pneumonia up to, but not including, Day 22 in the MITT Population. For the primary analysis, whether the subject has or has not developed *S. aureus* pneumonia will be based on sponsor defined outcome (SDO1).

The primary analysis is based on comparing two proportions of subjects who develop *S. aureus* pneumonia by SDO1 up to, but not including, Day 22. For each arm, the empirical proportion is defined by a ratio, which is the number of *S. aureus* pneumonia events divided

25OCTOBER2018 

by the total number of subjects in the arm. The inference about the difference of two population rates is based on the empirical counterpart. Specifically, the point estimate, 95% confidence interval and p-value for the rate difference. If subjects discontinued from the study due to any cause prior to Day 22, it will be considered as not developing *S. aureus* pneumonia by SDO1 for the primary efficacy analysis.

#### 3.5.2. Additional Analyses for *S. aureus* Pneumonia

Analyses of the primary efficacy endpoint will also be performed based on the PP Populations.

The following additional analyses will be performed in the MITT and PP Populations:

- The primary efficacy analysis, based on comparing two proportions of subjects who develop *S. aureus* pneumonia by SDO2 up to, but not including, Day 22. If subjects discontinued from the study due to any cause prior to Day 22 it will be considered as not developing *S. aureus* pneumonia for this analysis by SDO2.
- The additional analysis is based on comparing two proportions of subjects who develop *S. aureus* pneumonia by SDO1 and SDO2 up to, but not including, Day 22. For each arm, the empirical proportion is defined by a ratio, which is the number of *S. aureus* pneumonia events divided by the total number of subjects in the arm. The inference about the difference of two population rates is based on the empirical counterpart. Specifically, the point estimate, 95% confidence interval and p-value for the rate difference. If subjects discontinued from the study due to any cause prior to Day 22, data will be analyzed both as assumed to have developed *S. aureus* pneumonia and not having developed *S. aureus* pneumonia by SDO1 and SDO2.
- The Kaplan-Meier analysis will be performed for the proportion of subjects who develop *S. aureus* pneumonia by Day 21 as determined by SDO1 and SDO2. The proportion of subjects who develop *S. aureus* pneumonia up to but not including Day 22 will be obtained from Kaplan-Meier estimates for each treatment group. The number and percentage of subjects who developed *S. aureus* pneumonia or were censored will be summarized. The Kaplan-Meier estimate of event rates evaluated at Day 21 and the corresponding 95% confidence intervals will be presented for each treatment group. Subjects who did not develop *S. aureus* pneumonia, discontinued from the study, or died prior to Day 22 will be considered censored. For the censored subjects, the last assessment date on which the subject did not develop *S. aureus* pneumonia based on the Investigator's assessment will be used as the date of censoring.
- The additional Kaplan-Meier analysis will be performed for the proportion of subjects who develop *S. aureus* pneumonia by Day 21 as determined by SDO1 and SDO2. The proportion of subjects who develop *S. aureus* pneumonia up to but not including Day 22 will be obtained from Kaplan-Meier estimates for each treatment group. The number and percentage of subjects who developed *S. aureus* pneumonia or were censored will be summarized. The Kaplan-Meier estimate of event rates evaluated at Day 21 and the corresponding 95% confidence intervals will be

25OCTOBER2018 

presented for each treatment group. Discontinuation from the study due to any cause up to but not including Day 22 will be considered as an 'Event'.

• The Kaplan-Meier analysis will be performed for the proportion of subjects who develop *S. aureus* pneumonia up to but not including Day 22 as determined by the Investigator's judgement and the Review Meeting's determination of *S. aureus* as a causative pneumonia pathogen.

The number and percentage of subjects with SDO1 and SDO2 of *S. aureus* pneumonia, no *S. aureus* pneumonia, indeterminate, and censored in each treatment group will be summarized descriptively.

#### 3.5.3. Secondary Efficacy Endpoints

Duration of mechanical ventilation and length of hospital ICU stay during the first 21 days post-randomization will be summarized descriptively and compared between treatment groups using a Wilcoxon rank sum test in the MITT and PP Populations.

The other secondary endpoint, 28-day all-cause mortality in the MITT and PP Population, will be descriptively summarized by treatment group. All-cause mortality rate at Day 28 based on Kaplan-Meier estimates along with the 95% confidence interval will also be presented for each treatment group. Subjects whose survival status are unknown due to early termination or who are lost to follow up will be censored at the last day the subject was known to be alive.

### 3.5.4. Exploratory Efficacy Endpoints

Exploratory efficacy endpoints include:

- Proportion of subjects in the MITT and PP Populations with a diagnosis of HABP
   >48 hours post-extubation up to, but not including, Day 22 in extubated subjects;
- Proportion of subjects in the MITT and PP Populations with development of VABP up to, but not including, Day 22;
- Incidence of all pneumonias (SDO1 and SDO2) up to, but not including, Day 22 in the MITT and PP Populations, data will be analyzed both as assumed to have developed pneumonia and not having developed pneumonia by SDO1 and SDO2;
- Incidence of all bacterial pneumonias (SDO1 and SDO2) up to, but not including, Day 22 in the MITT and PP Populations, data will be analyzed both as assumed to have developed bacterial pneumonia and not having developed bacterial pneumonia by SDO1 and SDO2;
- Incidence of other non-*S. aureus* pneumonias (SDO1 and SDO2) up to, but not including, Day 22 in the MITT and PP Populations, data will be analyzed both as assumed to have developed non-*S. aureus* pneumonia and not having developed non-*S. aureus* pneumonia by SDO1 and SDO2;
- Incidence of Gram negative pneumonias (SDO1 and SDO2) up to, but not including, Day 22 in the MITT and PP Populations, data will be analyzed both as

25OCTOBER2018 

assumed to have developed Gram negative pneumonia and not having developed Gram negative pneumonia by SDO1 and SDO2;

- Incidence of other *S. aureus* (Non-Pulmonary *S. aureus*) infections acquired up to, but not including, Day 22 in the MITT and PP Populations.
- Summary of all-cause mortality rate through entire study period (through Day 90) in the MITT and PP Populations.

All exploratory efficacy endpoints will be descriptively summarized by treatment group.

## 3.6. Subgroup Analyses

The following subgroups will be used for subgroup analyses for the primary efficacy endpoint in the MITT Population, i.e. whether the subject has or doesn't have of *S. aureus* pneumonia up to, but not including, Day 22 for both SDO1 and SDO2 populations.

- Corrected randomization stratification (Receipt or Non-Receipt of concomitant anti-staphylococcal antibiotics at the time of randomization that are potentially active against *S. aureus* pneumonia.)
- Type of ICU (e.g., SICU, MICU, Neuro ICU, Trauma ICU)
- Length of stay in the intensive care unit (ICU) post-treatment (<5, 5-12, >12-22, and >22 days)
- Reason for mechanical ventilation
- BMI categories:  $<25, 25 < 30, 30 < 35, and \ge 35$
- Age: <50, 50-<65, and >65
- Male vs. female
- Acute kidney injury defined by an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (*viz.*, 0.3 mg/dL increase if baseline ≥0.6 mg/dL and 50% increase if baseline is ≤0.6 mg/dL) within 48 hours from receipt of study drug
- Presence of renal disease at Baseline: serum creatinine <2 mg/dL and ≥2 mg/dl.

The subgroup analyses for all-cause mortality rate at Day 28 and mortality rate through entire study period (through Day 90) will be performed by country in the MITT Population.

In addition, duration of mechanical ventilation and length of hospital ICU stay during the first 21 days post-randomization will be performed by the following subgroups in the MITT Population. Data will be analyzed both as assumed to have developed the following pneumonia and not having developed the following pneumonia by SDO1 and SDO2:

- All pneumonia (SDO1)
- All pneumonia (SDO2)
- S. aureus pneumonia (SDO1)
- *S. aureus* pneumonia (SDO2)

25OCTOBER2018 

- All bacterial pneumonia (SDO1)
- All bacterial pneumonia (SDO2)
- Non-S. aureus pneumonia (SDO1)
- Non-S. aureus pneumonia (SDO2)
- Gram negative pneumonia (SDO1)
- Gram negative pneumonia (SDO2)

## 3.7. Analysis of Safety Data

All subjects in the Safety Population will be included in the safety analyses and analyzed based on the actual treatment received.

#### 3.7.1. Adverse Events

Verbatim descriptions of Adverse Events (AEs) will be coded using Version 19.1 of MedDRA. Summary tables will be provided for all Treatment-Emergent Adverse Events (TEAEs). A TEAE is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration. All AEs (including non-TEAEs), Serious AEs (SAEs), and AEs leading to study drug discontinuation will be provided in listings by treatment group, subject ID, verbatim term, MedDRA system organ class (SOC) and preferred term (PT), start and end date, seriousness flag, severity, relationship to study drug, and action taken with study drug.

An overall summary of AEs will include the number and percentage of subjects in each treatment group who experienced at least one AE/TEAE in the following categories: any AE, any TEAE, any drug-related TEAE, any severe TEAE, any SAE, any drug-related SAE, any SAE leading to death, any TEAE leading to discontinuation of study drug, and any SAE leading to study drug discontinuation. Subjects with multiple events will be counted only once within each category. Severity grade and relationship will be counted using the maximum severity and the strongest relationship respectively for a subject with multiple TEAEs.

The number and percentage of subjects reporting a TEAE in each treatment group will be tabulated by SOC and PT; by SOC, PT, and severity; and by SOC, PT, and relationship (unrelated or related to study drug). For all analyses of TEAEs, if the same AE (based on PT) is reported for the same subject more than once, the AE is counted only once for that PT and at the highest severity and strongest relationship to study drug.

The number and percentage of subjects reporting a treatment-emergent SAE in each treatment group will be summarized by SOC and PT.

Listings will be provided for SAEs and AEs leading to drug discontinuation. In addition, all AEs will be listed.

25OCTOBER2018 

#### 3.7.2. Vital Signs

Vital sign measurements will include temperature, systolic and diastolic blood pressure, pulse, respiratory rate, and oxygenation status (as measured by pulse oximetry or arterial blood gas).

Descriptive statistics will be used to summarize vital signs measurements and change from baseline by each scheduled time point.

All vital sign assessments will be listed by subject.

#### 3.7.3. Clinical Laboratory Tests

Descriptive statistics will be provided for hematology, chemistry, urinalysis, and coagulation parameters and change from baseline by each scheduled time point.

Shift tables from baseline to the worst post-baseline value will be provided for selected chemistry parameters (Alanine aminotransferase, Aspartate aminotransferase, Total Bilirubin, Creatinine, and Alkaline phosphatase) and hematology parameters (Hematocrit, Hemoglobin, Platelets, White blood cell count and differential). Both scheduled and unscheduled visits will be considered. For chemistry parameters, the following categories will be used:  $\langle LLN, normal, \rangle ULN$  and  $\langle 3 \rangle ULN, \rangle 3 \rangle ULN$  to  $\langle 5 \rangle ULN, \rangle 5 \rangle ULN$ , and missing. For hematology parameters, the following categories will be used: low, normal, high, and missing.

The number and percentage of subjects with the following PCS abnormal liver function test will be summarized:

- ALT  $\ge 3 \times ULN$  and  $\ge 5 \times ULN$
- AST  $\geq 3 \times ULN$  and  $\geq 5 \times ULN$
- ALT or AST  $\ge 3 \times ULN$  and  $\ge 5 \times ULN$
- Total bilirubin  $\ge 1.5 \times ULN$  and  $\ge 2 \times ULN$
- ALP  $\geq$ 1.5×ULN and  $\geq$ 3×ULN
- ALT or AST  $\ge 3 \times ULN$  and Total bilirubin  $\ge 2 \times ULN$
- Potential Hy's Law cases: ALT or AST  $\ge 3 \times ULN$ , Total bilirubin  $\ge 2 \times ULN$ , and ALP  $\le 2 \times ULN$

A listing of subjects with any post-baseline abnormal liver function tests will be presented. All clinical laboratory data will be listed. Values outside the normal ranges will be flagged.

25OCTOBER2018 

## 4. GENERAL INFORMATION

#### 4.1. Statistical Software

The creation of analysis datasets and statistical analyses will be done using SAS® version 9.3 or higher. The Medpace standard operating procedures (Medpace documents GL-DS-02-S2.1 and GL-DS-03-S1) will be followed for the validation of all SAS programs and outputs.

# 4.2. Format of Tables, Listings, and Figures

The format of tables, listings, and figures will be described in a stand-alone programming specifications document and will be finalized before database lock for the study.

25OCTOBER2018 

# 5. APPENDIX

25OCTOBER2018 

# **Table Mock-Ups**

| TABLE 14.1.1.1 | 33 |
|---|---|
| Subject Disposition | |
| Intent-to-Treat Population | |
| TABLE 14.1.1.2 | 35 |
| Analysis Populations | |
| Intent-to-Treat Population | |
| TABLE 14.1.2.1 | 36 |
| Summary of Demographic and Baseline Characteristics | |
| Intent-to-Treat Population | |
| TABLE 14.1.2.2 | 41 |
| Summary of Demographic and Baseline Characteristics | |
| Modified Intent-to-Treat Population | |
| TABLE 14.1.2.3 | 41 |
| Summary of Demographic and Baseline Characteristics | |
| Per Protocol Population | |
| TABLE 14.1.2.4 | 41 |
| Summary of Demographic and Baseline Characteristics | |
| Safety Population | |
| TABLE 14.1.3 | 42 |
| Summary of Concomitant Medications | |
| Intent-to-Treat Population | |
| TABLE 14.2.1.1 | 43 |
| Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 | |
| Modified Intent-to-Treat Population | |
| TABLE 14.2.1.2 | 44 |
| Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 | |
| Per Protocol Population | |

| TABLE 14.2.1.3 |
|---|
| Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.1.4 |
| Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.1.5 |
| Additional Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But<br>Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.1.6 |
| Additional Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But<br>Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.1.7 |
| Additional Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But<br>Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.1.8 |
| Additional Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But<br>Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.2.1 |
| Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to<br>But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.2.2 |
| Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Per Protocol Population |

25OCTOBER2018 

| TABLE 14.2.2.3 |
|---|
| Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to<br>But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.2.4 |
| Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to<br>But Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.2.5 |
| Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.2.6 |
| Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.2.7 |
| Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.2.8 |
| Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Per Protocol Population |
| TABLE 14.2.2.9 |
| Kaplan-Meier Analysis of S. aureus Pneumonia Up to But Not Including Day 22 |
| Determined by Investigator's Judgement of S. aureus as a Causative Pneumonia Pathogen |
| Modified Intent-to-Treat Population |
| TABLE 14.2.2.10 |
| Kaplan-Meier Analysis of S. aureus Pneumonia Up to But Not Including Day 22 |
| Determined by Investigator's Judgement of S. aureus as a Causative Pneumonia Pathogen |
| Per Protocol Population |

25OCTOBER2018 

| TABLE 14.2.3.1.1 |
|---|
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Corrected Randomization Stratification |
| TABLE 14.2.3.1.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Corrected Randomization Stratification |
| TABLE 14.2.3.2.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Type of ICU at Baseline |
| TABLE 14.2.3.2.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Type of ICU at Baseline |
| TABLE 14.2.3.3.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Length of Stay in ICU Post-Treatment |
| TABLE 14.2.3.3.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Length of Stay in ICU Post-Treatment |

25OCTOBER2018 

| TABLE 14.2.3.4.1 |
|---|
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Baseline BMI Category |
| TABLE 14.2.3.4.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Baseline BMI Category |
| TABLE 14.2.3.5.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Age Group |
| TABLE 14.2.3.5.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Age Group |
| TABLE 14.2.3.6.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Gender |
| TABLE 14.2.3.6.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Gender |

25OCTOBER2018 

| TABLE 14.2.3.7.1 |
|---|
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Acute Kidney Injury Status within 48 hours from receipt of study drug |
| TABLE 14.2.3.7.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Acute Kidney Injury Status within 48 hours from receipt of study drug |
| TABLE 14.2.3.8.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Baseline Creatinine Category |
| TABLE 14.2.3.8.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Baseline Creatinine Category |
| TABLE 14.2.3.9.1 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Reason for Mechanical Ventilation at Baseline |
| TABLE 14.2.3.9.2 |
| Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia<br>Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| By Reason for Mechanical Ventilation at Baseline |
| TABLE 14.2.4.1.161 |
| Summary of Pneumonia Infection Rate Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |

25OCTOBER2018 

| TABLE 14.2.4.1.2 | 62 |
|---|---|
| Additional Summary of Pneumonia Infection Rate Up to But Not Including Day 22 | |
| Modified Intent-to-Treat Population | |
| TABLE 14.2.4.2.1 | 63 |
| Summary of Pneumonias Infection Rates Up to But Not Including Day 22 | |
| Per Protocol Population | |
| TABLE 14.2.4.2.2 | 63 |
| Additional Summary of Pneumonias Infection Rates Up to But Not Including Day 22 | |
| Per Protocol Population | |
| TABLE 14.2.5.1 | 64 |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization | |
| Modified Intent-to-Treat Population | |
| TABLE 14.2.5.2 | 65 |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization | |
| Per Protocol Population | |
| TABLE 14.2.5.3.1A | 66 |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO1) | |
| TABLE 14.2.5.3.1B | 67 |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Day<br>Post-Randomization | /S |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO1) | |
| TABLE 14.2.5.3.2A | 68 |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO2) | |

25OCTOBER2018 

| TABLE 14.2.5.3.2B |
|---|
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Pneumonia (SDO2) |
| TABLE 14.2.5.4.1A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with S. aureus Pneumonia (SDO1) |
| TABLE 14.2.5.4.1B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with S. aureus Pneumonia (SDO1) |
| TABLE 14.2.5.4.2A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with S. aureus Pneumonia (SDO2) |
| TABLE 14.2.5.4.2B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with S. aureus Pneumonia (SDO2) |
| TABLE 14.2.5.5.1A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO1) |

25OCTOBER2018 

| TABLE 14.2.5.5.1B |
|---|
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO1) |
| TABLE 14.2.5.5.2A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO2) |
| TABLE 14.2.5.5.2B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial pneumonia (SDO2) |
| TABLE 14.2.5.6.1A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S. aureus Pneumonia (SDO1) |
| TABLE 14.2.5.6.1B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S. aureus Pneumonia (SDO1) |
| TABLE 14.2.5.6.2A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S. aureus Pneumonia (SDO2) |

25OCTOBER2018 

| TABLE 14.2.5.6.2B |
|---|
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S. aureus Pneumonia (SDO2) |
| TABLE 14.2.5.7.1A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Gram Negative Pneumonia (SDO1) |
| TABLE 14.2.5.7.1B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Gram Negative Pneumonia (SDO1) |
| TABLE 14.2.5.7.2A |
| Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-<br>Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Gram Negative Pneumonia (SDO2) |
| TABLE 14.2.5.7.2B |
| Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Gram Negative Pneumonia (SDO2) |
| TABLE 14.2.6.1 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| TABLE 14.2.6.2 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Per Protocol Population |

25OCTOBER2018 

| TABLE 14.2.6.3.1A | 72 |
|---|---|
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO1) | |
| TABLE 14.2.6.3.1B | 73 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO1) | |
| TABLE 14.2.6.3.2A | 74 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO2) | |
| TABLE 14.2.6.3.2B | 74 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with All Pneumonia (SDO2) | |
| TABLE 14.2.6.4.1A | 74 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with S. aureus Pneumonia (SDO1) | |
| TABLE 14.2.6.4.1B | 74 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with S. aureus Pneumonia (SDO1) | |
| TABLE 14.2.6.4.2A | 74 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with S. aureus Pneumonia (SDO2) | |

25OCTOBER2018 

| TABLE 14.2.6.4.2B |
|---|
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with S. aureus Pneumonia (SDO2) |
| TABLE 14.2.6.5.1A |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO1) |
| TABLE 14.2.6.5.1B |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO1) |
| TABLE 14.2.5.6.2A |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial Pneumonia (SDO2) |
| TABLE 14.2.5.6.2B |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with All Bacterial pneumonia (SDO2) |
| TABLE 14.2.6.6.1A |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S. aureus Pneumonia (SDO1) |
| TABLE 14.2.6.6.1B |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization |
| Modified Intent-to-Treat Population |
| Subjects with Non-S, aureus Pneumonia (SDO1) |

25OCTOBER2018 


| TABLE 14.2.6.6.2A | 75 |
|---|---|
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Non-S. aureus Pneumonia (SDO2) | |
| TABLE 14.2.6.6.2B | 75 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Non-S. aureus Pneumonia (SDO2) | |
| TABLE 14.2.6.7.1A | 75 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Gram Negative Pneumonia (SDO1) | |
| TABLE 14.2.6.7.1B | 75 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Gram Negative Pneumonia (SDO1) | |
| TABLE 14.2.6.7.2A | 75 |
| Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Gram Negative Pneumonia (SDO2) | |
| TABLE 14.2.6.7.2B | 75 |
| Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization | |
| Modified Intent-to-Treat Population | |
| Subjects with Gram Negative Pneumonia (SDO2) | |
| TABLE 14.2.7.1 | 76 |
| Analysis of 28-Day All-Cause Mortality Rate | |
| Modified Intent-to-Treat Population | |
| TABLE 14.2.7.2 | 77 |
| Analysis of 28-Day All-Cause Mortality Rate | |
| Per Protocol Population | |

25OCTOBER2018

| TABLE 14.2.7.3 |
|---|
| Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90) |
| Modified Intent-to-Treat Population |
| TABLE 14.2.7.4 |
| Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90) |
| Per Protocol Population |
| TABLE 14.2.7.5 |
| Subgroup Analysis: Analysis of 28-Day All-Cause Mortality Rate |
| Modified Intent-to-Treat Population |
| By Country |
| TABLE 14.2.7.6 |
| Subgroup Analysis: Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90) |
| Modified Intent-to-Treat Population |
| By Country |
| TABLE 14.2.8.1 |
| Summary of Proportion of Subjects with Diagnosis of HABP >48 Hours Post-extubation Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| Extubated Subjects |
| TABLE 14.2.8.2 |
| Summary of Proportion of Subjects with Diagnosis of HABP >48 Hours Post-extubation Up to But Not Including Day 22 |
| Per Protocol Population |
| Extubated Subjects |
| TABLE 14.2.9.1 |
| Summary of Proportion of Subjects with Development of VABP Up to But Not Including Day 22 |
| Modified Intent-to-Treat Population |
| TABLE 14.2.9.2 |
| Summary of Proportion of Subjects with Development of VABP Up to But Not Including Day 22 |
| Per Protocol Population |

 25OCTOBER2018

| TABLE 14.3.1.1 | 84 |
|----------------------------------------------------------------------|----|
| Overview of Adverse Events | |
| Safety Population | |
| TABLE 14.3.1.2 | 85 |
| Subjects with Treatment-Emergent Adverse Events (TEAEs) | |
| By System Organ Class and Preferred Term | |
| Safety Population | |
| TABLE 14.3.1.3 | 86 |
| Subjects with Treatment-Emergent Serious Adverse Events (TESAEs) | |
| By System Organ Class and Preferred Term | |
| Safety Population | |
| TABLE 14.3.1.4 | 86 |
| Subjects with Drug-Related Treatment-Emergent Adverse Events | |
| By System Organ Class and Preferred Term | |
| Safety Population | |
| TABLE 14.3.1.5 | 87 |
| Subjects with Treatment-Emergent Adverse Events (TEAEs) | |
| By System Organ Class, Preferred Term and Maximum Severity | |
| Safety Population | |
| TABLE 14.3.1.6 | 88 |
| Subjects with Treatment-Emergent Adverse Events (TEAEs) | |
| By System Organ Class, Preferred Term and Relationship to Study Drug | |
| Safety Population | |
| TABLE 14.3.2.1 | 89 |
| Listing of Serious Adverse Events | |
| Safety Population | |
| TABLE 14.3.2.2 | 90 |
| Listing of Adverse Events Leading to Discontinuation of Study Drug | |
| Safety Population | |
| TABLE 14.3.3.1 | 91 |
| Summary of Laboratory Chemistry Parameters | |
| Safety Population | |

25OCTOBER2018

| TABLE 14.3.3.292 |
|---|
| Summary of Laboratory Hematology Parameters |
| Safety Population |
| TABLE 14.3.3.3 |
| Summary of Laboratory Coagulation Parameters |
| Safety Population |
| TABLE 14.3.3.4 |
| Summary of Laboratory Urinalysis Parameters |
| Safety Population |
| TABLE 14.3.3.593 |
| Shift Table for Hematology Parameters |
| Safety Population |
| TABLE 14.3.3.694 |
| Shift Table for Chemistry Parameters |
| Safety Population |
| TABLE 14.3.3.795 |
| Number (%) of Subjects with Prespecified Potentially Clinically Significant Abnormal Post-<br>Baseline Liver Function Tests |
| Safety Population |
| TABLE 14.3.3.8 |
| Listing of Subjects with Prespecified Potentially Clinically Significant Abnormal Post-<br>Baseline Liver Function Findings |
| Safety Population |
| TABLE 14.3.4 |
| Summary of Vital Signs |
| Safety Population |

25OCTOBER2018 

Arsanis, Inc.
Protocol No. ASN100-201

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

# Table 14.1.1.1 Subject Disposition Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) | Total<br>(N=###)<br>n (%) |
|---|---|---|---|
| Subjects who randomized in primary prevention study | ### (###.#) | ### (###.#) | ### (###.#) |
| Subjects who randomized in treatment sub-study [1] | ### (###.#) | ### (###.#) | ### (###.#) |
| Subjects who received study drug | ### (###.#) | ### (###.#) | ### (###.#) |
| Subjects who completed the study assessments through Day 22 | ### (###.#) | ### (###.#) | ### (###.#) |
| Subjects who did not complete the study assessments through Day 22 | ### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018 

<sup>[1]</sup> A single subject 268-002-118 was enrolled and randomized into the treatment sub-study. This subject is only included in tabulations presenting disposition and safety data.


Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.1.1.1 Subject Disposition Intent-to-Treat Population Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

| | ASN100 | | | | Total | |
|---|---|---|---|---|---|---|
| | • | (%) | | =###)<br>(왕) | | (%) |
| ubjects who completed the study assessments through Day 90 | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| subjects who did not complete the study assessments through Day 90 | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Adverse event | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Death | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Lost to follow-up | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Non-compliance with study drug | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Physician decision | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Protocol deviation | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Withdrawal of consent by LAR | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Withdrawal of consent by subject | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Discontinuation by subject | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Discontinuation by LAR | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| Other | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| subjects who completed assessments through Day 22, but did not complete the study assessments through Day 90 | ### | (###.#) | ### | (###.#) | ### | (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018 

<sup>[1]</sup> A single subject 268-002-118 was enrolled and randomized into the treatment sub-study. This subject is only included in tabulations presenting disposition and safety data.

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

# Table 14.1.1.2 Analysis Populations Intent-to-Treat Population

| | ASN100 | Placebo | Total |
|---|---|---|---|
| | (N=###) | (N=###) | (N=###) |
| | n (%) | n (%) | n (%) |
| Intent-to-Treat (ITT) Population [1] | ### (###.#) | ### (###.#) | ### (###.#) |
| Modified Intent-to-Treat (MITT) Population [2] | ### (###.#) | ### (###.#) | ### (###.#) |
| Per Protocol (PP) Population [3] | ### (###.#) | ### (###.#) | ### (###.#) |
| Safety Population [4] | ### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

- [1] Intent-to-Treat Population includes all subjects who are randomized to receive study drug.
- [2] Modified Intent-to-Treat Population includes subjects in the ITT Population who receive study drug and who are heavily colonized with S. aureus as determined by quantitative or semi-quantitative culture of an ETA specimen.
- [3] Per Protocol Population includes all subjects in the MITT Population who also meet the criteria specified in the SAP.
- [4] Safety Population includes all subjects who receive any amount of study drug and have at least 1 post-treatment safety assessment.

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.1.2.1

Summary of Demographic and Baseline Characteristics
Intent-to-Treat Population

| Demographics/Characteristics<br>Category/Statistic | ASN100<br>(N=###) | Placebo (N=###) | Total<br>(N=###) |
|---|---|---|---|
| Age (years) | | | |
| n | ### | ### | ### |
| Mean | ##.# | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## | ##.## |
| Minimum | ## | ## | ## |
| Median | ##.# | ##.# | ##.# |
| Maximum | ## | ## | ## |
| Age group 1 (n, %) | | | |
| <55 years | ### (###.#) | ### (###.#) | ### (###.#) |
| 55 - <65 years | ### (###.#) | ### (###.#) | ### (###.#) |
| 65 - <75 years | ### (###.#) | ### (###.#) | ### (###.#) |
| >=75 years | ### (###.#) | ### (###.#) | ### (###.#) |
| age group 2 (n, %) | | | |
| <50 years | ### (###.#) | ### (###.#) | ### (###.#) |
| 50 - <65 years | ### (###.#) | ### (###.#) | ### (###.#) |
| >=65 years | ### (###.#) | ### (###.#) | ### (###.#) |
| Gender (n, %) | | | |
| Male | ### (###.#) | ### (###.#) | ### (###.#) |
| Female | ### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018 

<sup>[1]</sup> Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL Increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.
Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


# Table 14.1.2.1 Summary of Demographic and Baseline Characteristics Intent-to-Treat Population

| Demographics/Characteristics<br>Category/Statistic | ASN100<br>(N=###) | Placebo<br>(N=###) | Total<br>(N=###) |
|---|---|---|---|
| Race (n, %) | | | |
| American Indian or Alaska Native | ### (###.#) | ### (###.#) | ### (###.#) |
| Asian | ### (###.#) | ### (###.#) | ### (###.#) |
| Black or African American | ### (###.#) | ### (###.#) | ### (###.#) |
| Native Hawaiian or other Pacific Islander | ### (###.#) | ### (###.#) | ### (###.#) |
| White | ### (###.#) | ### (###.#) | ### (###.#) |
| Other | ### (###.#) | ### (###.#) | ### (###.#) |
| Tthnicity (n, %) | | | |
| Hispanic or Latino | ### (###.#) | ### (###.#) | ### (###.#) |
| Not Hispanic or Latino | ### (###.#) | ### (###.#) | ### (###.#) |
| Not reported | ### (###.#) | ### (###.#) | ### (###.#) |
| Unknown | ### (###.#) | ### (###.#) | ### (###.#) |
| Jeight (kg) | | | |
| n | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## |
| Standard Deviation | ##.## | ##.## | ##.## |
| Minimum | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ## - # |
| Height (cm) | | | |
| n | ### | ### | ### |
| Mean | ##.# | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## | ##.## |
| Minimum | ## | ## | ## |
| Median | ##.# | ##.# | ##.# |
| Maximum | ## | ## | ## |

Percentage is calculated using the number of subjects in the column heading as the denominator. Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018 

<sup>[1]</sup> Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL Increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


## Table 14.1.2.1 Summary of Demographic and Baseline Characteristics Intent-to-Treat Population

| Demographics/Characteristics | ASN100 | Placebo | Total |
|---|---|---|---|
| Category/Statistic | (N=###) | (N=###) | (N=##) |
| Body Mass Index (kg/m^2) | | | |
| n | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## |
| Standard Deviation | ##.### | ##.## | ##.## |
| Minimum | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# |
| Body Mass Index category (n, %) | | | |
| <25 kg/m^2 | ### (###.#) | ### (###.#) | ### (###.#) |
| 25-<30 kg/m^2 | ### (###.#) | ### (###.#) | ### (###.#) |
| 30-<35 kg/m^2 | ### (###.#) | ### (###.#) | ### (###.#) |
| >=35 kg/m^2 | ### (###.#) | ### (###.#) | ### (###.#) |
| Corrected randomization stratification (Recei | nt of concemitant anti-stanbuloss | agaal antihiotiga at | time of randomization |
| that are potentially active against S. aure | | occar ancibiocics at | cline of fandomization |
| Yes | ### (###.#) | ### (###.#) | ### (###.#) |
| No | ### (###.#) | ### (###.#) | ### (###.#) |
| | """ ("""•") | """ (""", | " " " ( " " " ) |
| Type of Hospital Unit at Time of ICF (n, %) | | | |
| ICU | ### (###.#) | ### (###.#) | ### (###.#) |
| MICU - Medical ICU | ### (###.#) | ### (###.#) | ### (###.#) |
| SICU - Surgical ICU | ### (###.#) | ### (###.#) | ### (###.#) |
| TICU - Trauma ICU | ### (###.#) | ### (###.#) | ### (###.#) |
| 377.077 37 7.077 | ### (###.#) | ### (###.#) | ### (###.#) |
| NICU - Neuro ICU | | 0.00 / 0.00 0.5 | |
| NICU - Neuro ICU<br>CCU - Coronary Care Unit | ### (###.#) | ### (###.#) | ### (###.#) |
| | ### (###.#)<br>### (###.#) | ### (###.#)<br>### (###.#) | ### (###.#)<br>### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018 

<sup>[1]</sup> Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL Increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


# Table 14.1.2.1 Summary of Demographic and Baseline Characteristics Intent-to-Treat Population

| emographics/Characteristics<br>Category/Statistic | ASN100<br>(N=###) | Placebo<br>(N=###) | Total<br>(N=###) |
|---|---|---|---|
| Category/Statistic | (IV—###) | (N-###) | (14-###) |
| ength of stay (total days) in ICU post-treatment | | | |
| n | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## |
| Standard Deviation | ##.## | ##.## | ##.## |
| Minimum | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# |
| ength of stay in ICU post-treatment category (n, %) | | | |
| <5 days | ### (###.#) | ### (###.#) | ### (###.#) |
| 5-12 days | ### (###.#) | ### (###.#) | ### (###.#) |
| >12-22 days | ### (###.#) | ### (###.#) | ### (###.#) |
| >22 days | ### (###.#) | ### (###.#) | ### (###.#) |
| cute kidney injury status at Day 2 visit (n, %) [1] | | | |
| Yes | ### (###.#) | ### (###.#) | ### (###.#) |
| No | ### (###.#) | ### (###.#) | ### (###.#) |
| aseline creatinine (mg/dL) | | | |
| n | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## |
| Standard Deviation | ##.### | ##.### | ##.### |
| Minimum | ##.## | ##.## | ##.## |
| Median | ##.## | ##.## | ##.## |
| Maximum | ##.## | ##.## | ##.## |
| aseline creatinine category (n, %) | | | |
| <2 mg/dL | ### (###.#) | ### (###.#) | ### (###.#) |
| >=2 mg/dL | ### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018 

<sup>[1]</sup> Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL Increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


# Table 14.1.2.1 Summary of Demographic and Baseline Characteristics Intent-to-Treat Population

| Demographics/Characteristics<br>Category/Statistic | ASN100<br>(N=###) | Placebo (N=###) | Total (N=###) |
|---|---|---|---|
| eason for mechanical ventilation at baseline (n. | , %) | | |
| Cardiovascular impairment | ### (###.#) | ### (###.#) | ### (###.#) |
| · · | • | ### (###.#)<br>### (###.#) | ### (###.#)<br>### (###.#) |
| Cardiovascular impairment | ### (###.#) | | |
| Cardiovascular impairment<br>Neurological impairment | ### (###.#)<br>### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018 

<sup>[1]</sup> Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL Increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.

The layouts of the following tables will be the same as Table 14.1.2.1:

Table 14.1.2.2

Summary of Demographic and Baseline Characteristics Modified Intent-to-Treat Population

Table 14.1.2.3

Summary of Demographic and Baseline Characteristics Per Protocol Population

Table 14.1.2.4

Summary of Demographic and Baseline Characteristics  ${\tt Safety\ Population}$ 

25OCTOBER2018 

Arsanis, Inc.


Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

### Table 14.1.3 Summary of Concomitant Medications Intent-to-Treat Population

| ATC Classification Preferred Term | ASN100 | Placebo | Total |
|---|---|---|---|
| | (N=###) | (N=###) | (N=###) |
| | n (%) | n (%) | n (%) |
| Any concomitant medications | ### (###.#) | ### (###.#) | ### (###.#) |
| ATC Classification 1 Preferred Term 1 Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |
| | ### (###.#) | ### (###.#) | ### (###.#) |
| | ### (###.#) | ### (###.#) | ### (###.#) |
| ATC Classification 2 Preferred Term 1 Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |
| | ### (###.#) | ### (###.#) | ### (###.#) |
| | ### (###.#) | ### (###.#) | ### (###.#) |

Coding is based on WHO Drug Dictionary Sept 2016E.

Percentage is calculated using the number of subjects in the column heading as the denominator.

Concomitant medications are medications used on or after the initiation of study drug administration.

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

#### Table 14.2.1.1

Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###) | Placebo (N=###) | Treati | ment Comparison [1] | |
|---|---|---|---|---|---|
| SDO1 | n (%) | n (%) | Difference (%) | 95% CI | P-value |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.#### |
| No | ### (###.#) | ### (###.#) | ππ•π | (##•##, ##•#) | #•### |
| Censored | ### (###.#) | ### (###.#) | | | |
| Indeterminate | ### (###.#) | ### (###.#) | | | |

Percentage is calculated using the number of subjects in the column heading as the denominator.

[1] Treatment difference (ASN100 - Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO1 between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.

Note: In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing S. aureus pneumonia.

25OCTOBER2018 

The layout of the following table will be the same as Table 14.2.1.1:

Table 14.2.1.2

Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Table 14.2.1.3

Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###) | Placebo<br>(N=###) | Treat: | ment Comparison [1] | |
|---|---|---|---|---|---|
| SDO2 | n (%) | n (%) | Difference (%) | 95% CI | P-value |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.#### |
| No | ### (###.#) | ### (###.#) | " " • " | ( - | " • " " " |
| Censored | ### (###.#) | ### (###.#) | | | |
| Indeterminate | ### (###.#) | ### (###.#) | | | |

Percentage is calculated using the number of subjects in the column heading as the denominator.

[1] Treatment difference (ASN100 - Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO2 between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.

Note: In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing S. aureus pneumonia.

25OCTOBER2018 

The layout of the following table will be the same as Table 14.2.1.3:

Table 14.2.1.4

Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.1.5

Additional Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###) | Placebo<br>(N=###) | | ment Comparison [1] | |
|---|---|---|---|---|---|
| Category | n (%) | n (%) | Difference (%) | 95% CI | P-value |
| SD01=Yes + Presumed S. aureus Pneumonia [2] | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.### |
| SD01=Yes | ### (###.#) | ### (###.#) | | | |
| Presumed S. aureus Pneumonia [2] | ### (###.#) | ### (###.#) | | | |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018 

<sup>[1]</sup> Treatment difference (ASN100 - Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO1 and Presumed S. aureus pneumonia between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.

<sup>[2]</sup> In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as developing S. aureus pneumonia, i.e., Presumed S. aureus pneumonia.

The layout of the following table will be the same as Table 14.2.1.5:

Table 14.2.1.6

Additional Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.1.7

Additional Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###) | Placebo<br>(N=###) | Treat | ment Comparison [1] | |
|---|---|---|---|---|---|
| Category | n (%) | n (%) | Difference (%) | 95% CI | P-value |
| SDO2=Yes + Presumed S. aureus Pneumonia [2] | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.### |
| SDO2=Yes | ### (###.#) | ### (###.#) | | | |
| Presumed S. aureus Pneumonia [2] | ### (###.#) | ### (###.#) | | | |

Percentage is calculated using the number of subjects in the column heading as the denominator.

- [1] Treatment difference (ASN100 Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO2 and Presumed S. aureus pneumonia between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.
- [2] In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as developing S. aureus pneumonia, i.e., Presumed S. aureus pneumonia.

25OCTOBER2018 

The layout of the following table will be the same as Table 14.2.1.7:

Table 14.2.1.8

Additional Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

25OCTOBER2018 

Addendum to SAP, Version 1.0

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.2.1

Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| Subjects with S. aureus pneumonia up to but not including Day 22 | ### (###.#) | ### (###.#) |
| Subjects censored | ### (###.#) | ### (###.#) |
| Kaplan-Meier Estimate (95% CI) | ##.# (##.#, ##.#) | ##.# (##.#, ##.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

Note: Subjects who did not develop S. aureus pneumonia, discontinued from the study, or died prior to Day 22 will be considered censored.

25OCTOBER2018 

## The layouts of the following tables will be the same as Table 14.2.2.1:

Table 14.2.2.2

Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

Table 14.2.2.3

Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Modified Intent-to-Treat Population

Table 14.2.2.4

Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.
Protocol Number: ASN100-201


Table 14.2.2.5

Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Modified Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| Subjects with S. aureus pneumonia up to but not including Day 22 | ### (###.#) | ### (###.#) |
| Subjects censored | ### (###.#) | ### (###.#) |
| Kaplan-Meier Estimate (95% CI) | ##.# (##.#, ##.#) | ##.# (##.#, ##.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Note: Discontinuation from the study due to any cause up to but not including Day 22 will be considered as an event.

25OCTOBER2018 

## The layouts of the following tables will be the same as Table 14.2.2.5:

Table 14.2.2.6

Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

Table 14.2.2.7

Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Modified Intent-to-Treat Population

Table 14.2.2.8

Additional Kaplan-Meier Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.2.9

Kaplan-Meier Analysis of S. aureus Pneumonia Up to But Not Including Day 22 Determined by Investigator's Judgement of S. aureus as a Causative Pneumonia Pathogen Modified Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| Subjects with S. aureus pneumonia up to but not including Day 22 | ### (###.#) | ### (###.#) |
| Subjects censored | ### (###.#) | ### (###.#) |
| Kaplan-Meier Estimate (95% CI) | ##.# (##.#, ##.#) | ##.# (##.#, ##.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Determination of S. aureus as causative pathogen was confirmed and accepted by Sponsor at review meeting.

25OCTOBER2018 

The layouts of the following tables will be the same as Table 14.2.2.9

Table 14.2.2.10

Kaplan-Meier Analysis of S. aureus Pneumonia Up to But Not Including Day 22 Determined by Investigator's Judgement of S. aureus as a Causative Pneumonia Pathogen Per Protocol Population

 25OCTOBER2018

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.
Protocol Number: ASN100-201


Table 14.2.3.1.1

Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22

Modified Intent-to-Treat Population

By Corrected Randomization Stratification

| Subgroup | ASN100 | Placebo | Treatme | nt Comparison [1] | |
|---|---|---|---|---|---|
| SDO1 | n/N' (%) | n/N' (%) | Difference (%) | 95% CI | P-value |
| eceipt of concomitant anti-sta | phylococcal antibiotics at the t: | ime of randomization | 1 | | |
| hat are potentially active aga | inst S. aureus pneumonia | | | | |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.### |
| No | ### (###.#) | ### (###.#) | | | |
| Censored | ### (###.#) | ### (###.#) | | | |
| Indeterminate | ### (###.#) | ### (###.#) | | | |
| Non-Receipt of concomitant anti | -staphylococcal antibiotics at the | ne time of randomiza | ation | | |
| that are potentially active aga | inst S. aureus pneumonia | | | | |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.#### |
| No | ### (###.#) | ### (###.#) | | | |
| 0 | ### (###.#) | ### (###.#) | | | |
| Censored | | | | | |

Percentage is calculated using N' which is the number of subjects in each subgroup as the denominator.

[1] Treatment difference (ASN100 - Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO1 at specified subgroup between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.

Note: In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing S. aureus pneumonia.

25OCTOBER2018 

Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.3.1.2

Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22

Modified Intent-to-Treat Population

By Corrected Randomization Stratification

| Subgroup | ASN100 | Placebo | Treatme | ent Comparison [1] | |
|---|---|---|---|---|---|
| SDO2 | n/N' (%) | n/N' (%) | Difference (%) | 95% CI | P-value |
| Receipt of concomitant anti-staphy | alogoggal antibiotics at the ti | mo of randomization | | | |
| that are potentially active agains | | .me or randomizacion | 1 | | |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.### |
| No | ### (###.#) | ### (###.#) | | , , , | |
| Censored | ### (###.#) | ### (###.#) | | | |
| Indeterminate | ### (###.#) | ### (###.#) | | | |
| Non-Receipt of concomitant anti-st | aphylococcal antibiotics at th | ne time of randomiza | ation | | |
| that are potentially active agains | | o cime of fanacmila | .01011 | | |
| Yes | ### (###.#) | ### (###.#) | ##.# | (##.##, ##.#) | #.#### |
| No | ### (###.#) | ### (###.#) | | , | |
| Censored | ### (###.#) | ### (###.#) | | | |

Percentage is calculated using N' which is the number of subjects in each subgroup as the denominator.

[1] Treatment difference (ASN100 - Placebo) is the estimate of the difference in the S. aureus pneumonias rate based on SDO2 at specified subgroup between the two treatment arms. The difference estimates, the 95% CIs, and P-values are obtained based on Wald test on equality of proportions.

Note: In subjects who are not confirmed as having S. aureus pneumonia and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing S. aureus pneumonia.

25OCTOBER2018 

```
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                             By Type of ICU at Baseline
                                                  Table 14.2.3.2.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                             By Type of ICU at Baseline
                                                  Table 14.2.3.3.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                      By Length of Stay in ICU Post-Treatment
                                                  Table 14.2.3.3.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                      By Length of Stay in ICU Post-Treatment
                                                  Table 14.2.3.4.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                              By Baseline BMI Category
                                                  Table 14.2.3.4.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                              By Baseline BMI Category
                                                  Table 14.2.3.5.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                                    By Age Group
                                                  Table 14.2.3.5.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                                    By Age Group
                                                  Table 14.2.3.6.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                                      By Gender
```

Table 14.2.3.6.2 Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22 Modified Intent-to-Treat Population By Gender

Addendum to SAP. Version 1.0

25OCTOBER2018 

### The layouts of the following tables will be the same as Tables 14.2.3.1.1 and 14.2.3.1.2:

<< Programing note: for tables 14.2.3.7.1 and 14.2.3.7.2, add footnote "Acute kidney injury is defined as an absolute increase in serum creatinine of 0.3 mg/dL or a 50% increase (i.e., 0.3 mg/dL increase if baseline >=0.6 mg/dL and 50% increase if baseline is <=0.6 mg/dL) within 48 hours from receipt of study drug.">>

```
Table 14.2.3.7.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                     By Acute Kidney Injury Status within 48 hours from receipt of study drug
                                                  Table 14.2.3.7.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                     By Acute Kidney Injury Status within 48 hours from receipt of study drug
                                                  Table 14.2.3.8.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                          By Baseline Creatinine Category
                                                  Table 14.2.3.8.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                          By Baseline Creatinine Category
                                                  Table 14.2.3.9.1
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO1) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                  By Reason for Mechanical Ventilation at Baseline
                                                  Table 14.2.3.9.2
Subgroup Analysis - Analysis of Sponsor-Defined Outcome (SDO2) of S. aureus Pneumonia Up to But Not Including Day 22
                                        Modified Intent-to-Treat Population
                                  By Reason for Mechanical Ventilation at Baseline
```

25OCTOBER2018 


Arsanis, Inc.
Protocol Number: ASN100-201

Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM
Table 14.2.4.1.1

Program Name: XXXX.sas

Table 14.2.4.1.1
Summary of Pneumonia Infection Rate Up to But Not Including Day 22
Modified Intent-to-Treat Population

| | ASN100 | Placebo |
|----------------------------------------|------------------|------------------|
| Category | (N=###)<br>n (%) | (N=###)<br>n (%) |
| | 11 (%) | 11 (%) |
| All pneumonia (SDO1) | ### (###.#) | ### (###.#) |
| All pneumonia (SDO2) | ### (###.#) | ### (###.#) |
| S. aureus pneumonia (SDO1) | ### (###.#) | ### (###.#) |
| S. aureus pneumonia (SDO2) | ### (###.#) | ### (###.#) |
| All bacterial pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| All bacterial pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Non-S. aureus pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| Non-S. aureus pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Gram negative pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| Gram negative pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Non-pulmonary S. aureus infection rate | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

Note: In subjects who are not confirmed as having the specific category and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing that category.

25OCTOBER2018 

Arsanis, Inc. Protocol Number: ASN100-201 

Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Addendum to SAP, Version 1.0

Table 14.2.4.1.2 Additional Summary of Pneumonia Infection Rate Up to But Not Including Day 22 Modified Intent-to-Treat Population

| Category | ASN100<br>(N=##)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| | 11 (*0) | 11 (0) |
| All pneumonia (SDO1) | ### (###.#) | ### (###.#) |
| All pneumonia (SDO2) | ### (###.#) | ### (###.#) |
| S. aureus pneumonia (SDO1) | ### (###.#) | ### (###.#) |
| S. aureus pneumonia (SDO2) | ### (###.#) | ### (###.#) |
| All bacterial pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| All bacterial pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Non-S. aureus pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| Non-S. aureus pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Gram negative pneumonia rate (SDO1) | ### (###.#) | ### (###.#) |
| Gram negative pneumonia rate (SDO2) | ### (###.#) | ### (###.#) |
| Non-pulmonary S. aureus infection rate | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator. Note: In subjects who are not confirmed as having the specific category and who are discontinued from the study due to any cause prior to Day 22, they are considered as developing that category.

25OCTOBER2018  The layouts of the following tables will be the same as Table 14.2.4.1.1 and 14.2.4.1.2:

Table 14.2.4.2.1

Summary of Pneumonias Infection Rates Up to But Not Including Day 22 Per Protocol Population

Table 14.2.4.2.2

Additional Summary of Pneumonias Infection Rates Up to But Not Including Day 22 Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.5.1

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=###) |
|--------------------|-------------------|--------------------|
| n | ## | ## |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

25OCTOBER2018 

Total duration (days) of mechanical ventilation is defined as total number of days on mechanical ventilation during the first 21 days post-randomization.

The layout of the following table will be the same as Table 14.2.5.1:

Table 14.2.5.2

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Per Protocol Population

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.2.5.3.1a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population Subjects with All Pneumonia (SDO1)

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=###) |
|--------------------|-------------------|--------------------|
| n | ## | ## |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

Total duration (days) of mechanical ventilation is defined as total number of days on mechanical ventilation during the first 21 days post-randomization.

Note: In subjects who are not confirmed as having pneumonia (SDO1) and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing pneumonia (SDO1).

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.2.5.3.1b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population Subjects with All Pneumonia (SDO1)

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=###) |
|--------------------|-------------------|--------------------|
| n | ## | ## |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

Total duration (days) of mechanical ventilation is defined as total number of days on mechanical ventilation during the first 21 days post-randomization.

Note: In subjects who are not confirmed as having pneumonia (SDO1) and who are discontinued from the study due to any cause prior to Day 22, they are considered as developing pneumonia (SDO1).

25OCTOBER2018 

### The layouts of the following tables will be the same as Table 14.2.5.3.1a and 14.2.5.3.1b:

Table 14.2.5.3.2a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Pneumonia (SDO2)

Table 14.2.5.3.2b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Pneumonia (SDO2)

Table 14.2.5.4.1a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO1)

Table 14.2.5.4.1b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO1)

Table 14.2.5.4.2a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO2)

Table 14.2.5.4.2b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO2)

Table 14.2.5.5.1a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO1)

Table 14.2.5.5.1b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO1)

Table 14.2.5.5.2a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO2)

25OCTOBER2018 

Table 14.2.5.5.2b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population

Subjects with All Bacterial pneumonia (SDO2)

Table 14.2.5.6.1a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO1)

Table 14.2.5.6.1b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO1)

Table 14.2.5.6.2a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO2)

Table 14.2.5.6.2b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO2)

Table 14.2.5.7.1a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Gram Negative Pneumonia (SDO1)

Table 14.2.5.7.1b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population Subjects with Gram Negative Pneumonia (SDO1)

Table 14.2.5.7.2a

Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Gram Negative Pneumonia (SDO2)

Table 14.2.5.7.2b

Additional Analysis of Total Duration (Days) of Mechanical Ventilation During First 21 Days Post-Randomization Subjects with Gram Negative Pneumonia (SDO2)

Modified Intent-to-Treat Population

25OCTOBER2018  Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

#### Table 14.2.6.1

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization  ${\tt Modified\ Intent-to-Treat\ Population}$ 

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=###) |
|--------------------|-------------------|--------------------|
| n | ## | ## |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

Total length of ICU stay (days) is defined as the total number of days of ICU stay during the first 21 days post-randomization.

25OCTOBER2018 

The layout of the following table will be the same as Table 14.2.6.1:

Table 14.2.6.2

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.6.3.1a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization Modified Intent-to-Treat Population Subjects with All Pneumonia (SDO1)

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=####) |
|--------------------|-------------------|---------------------|
| n | ### | ### |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

Total length of ICU stay (days) is defined as the total number of days of ICU stay during the first 21 days post-randomization. Note: In subjects who are not confirmed as having pneumonia (SDO1) and who are discontinued from the study due to any cause prior to Day 22, they are considered as not developing pneumonia (SDO1).

25OCTOBER2018 
Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.2.6.3.1b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization Modified Intent-to-Treat Population

Subjects with All Pneumonia (SDO1)

| Statistics | ASN100<br>(N=###) | Placebo<br>(N=###) |
|--------------------|-------------------|--------------------|
| n | ## | ## |
| Mean | ##.# | ##.# |
| Standard Deviation | ##.## | ##.## |
| Minimum | ## | ## |
| Median | ##.# | ##.# |
| Maximum | ## | ## |

<sup>[1]</sup> P-value is obtained from a Wilcoxon rank sum test.

25OCTOBER2018 

Total length of ICU stay (days) is defined as the total number of days of ICU stay during the first 21 days post-randomization. Note: In subjects who are not confirmed as having pneumonia (SDO1) and who are discontinued from the study due to any cause prior to Day 22, they are considered as developing pneumonia (SDO1).

#### The layouts of the following tables will be the same as Table 14.2.6.3.1a and 14.2.6.3.1b:

Table 14.2.6.3.2a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization
Modified Intent-to-Treat Population
Subjects with All Pneumonia (SDO2)

Table 14.2.6.3.2b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization Modified Intent-to-Treat Population Subjects with All Pneumonia (SDO2)

Table 14.2.6.4.1a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO1)

Table 14.2.6.4.1b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population
Subjects with S. aureus Pneumonia (SDO1)

Table 14.2.6.4.2a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with S. aureus Pneumonia (SDO2)

Table 14.2.6.4.2b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population
Subjects with S. aureus Pneumonia (SDO2)

Table 14.2.6.5.1a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO1)

Table 14.2.6.5.1b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO1)

Table 14.2.5.6.2a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial Pneumonia (SDO2)

25OCTOBER2018 

Table 14.2.5.6.2b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with All Bacterial pneumonia (SDO2)

Table 14.2.6.6.1a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization
Modified Intent-to-Treat Population
Subjects with Non-S. aureus Pneumonia (SDO1)

Table 14.2.6.6.1b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO1)

Table 14.2.6.6.2a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization
Modified Intent-to-Treat Population
Subjects with Non-S. aureus Pneumonia (SDO2)

Table 14.2.6.6.2b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Non-S. aureus Pneumonia (SDO2)

Table 14.2.6.7.1a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization
Modified Intent-to-Treat Population
Subjects with Gram Negative Pneumonia (SDO1)

Table 14.2.6.7.1b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Gram Negative Pneumonia (SDO1)

Table 14.2.6.7.2a

Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization
Modified Intent-to-Treat Population
Subjects with Gram Negative Pneumonia (SDO2)

Table 14.2.6.7.2b

Additional Analysis of Total Length of ICU Stay (Days) During First 21 Days Post-Randomization

Modified Intent-to-Treat Population

Subjects with Gram Negative Pneumonia (SDO2)

25OCTOBER2018 

Arsanis, Inc.

Addendum to SAP, Version 1.0

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

## Table 14.2.7.1 Analysis of 28-Day All-Cause Mortality Rate Modified Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| 28-Day all-cause mortality rate | ### (###.#) | ### (###.#) |
| Subjects censored | ### (###.#) | ### (###.#) |
| Kaplan-Meier Estimate (95% CI) | ##.# (##.#, ##.#) | ##.# (##.#, ##.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018 

The layouts of the following tables will be the same as Table 14.2.7.1:

Table 14.2.7.2

Analysis of 28-Day All-Cause Mortality Rate
Per Protocol Population

Table 14.2.7.3

Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90) Modified Intent-to-Treat Population

Table 14.2.7.4

Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90) Per Protocol Population

25OCTOBER2018 

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Table 14.2.7.5

Subgroup Analysis: Analysis of 28-Day All-Cause Mortality Rate
Modified Intent-to-Treat Population
By Country

| Subgroup | ASN100<br>(N=###)<br>n/N' (%) | Placebo<br>(N=###)<br>n/N' (%) |
|---|---|---|
| Country 1<br>28-Day all-cause mortality rate | ###/### (###.#) | ###/### (###.#) |
| Subjects censored | ###/### (###.#) | ###/### (###.#) |
| Kaplan-Meier Estimate (95% CI) | ###/### (###.#) | ###/### (###.#) |
| Country 2 | | |

Percentage is calculated using N' which is the number of subjects in each subgroup as the denominator.

25OCTOBER2018 

The layout of the following table will be the same as Table 14.2.7.5:

Table 14.2.7.6

Subgroup Analysis: Analysis of All-Cause Mortality Rate Through Entire Study Period (Through Day 90)

Modified Intent-to-Treat Population

By Country

25OCTOBER2018 


Arsanis, Inc. Protocol Number: ASN100-201

Run Date: MM/DD/YYYY HH:MM  Data Last Modified: MM/DD/YYYY HH:MM

Table 14.2.8.1

Summary of Proportion of Subjects with Diagnosis of HABP >48 Hours Post-extubation Up to But Not Including Day 22 Modified Intent-to-Treat Population Extubated Subjects

Program Name: XXXX.sas

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| Subjects with diagnosis of HABP >48 hours<br>Post-extubation up to but not including Day 22 | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018  The layout of the following table will be the same as Table 14.2.8.1:

Table 14.2.8.2

Summary of Proportion of Subjects with Diagnosis of HABP >48 Hours Post-extubation Up to But Not Including Day 22

Per Protocol Population

Extubated Subjects

25OCTOBER2018 


Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.2.9.1

Summary of Proportion of Subjects with Development of VABP Up to But Not Including Day 22 Modified Intent-to-Treat Population

| | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) |
|---|---|---|
| Subjects with development of VABP up to but not including Day 22 | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

25OCTOBER2018 

Per Protocol Population

The layout of the following table will be the same as Table 14.2.9.1:

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.3.1.1
Overview of Adverse Events
Safety Population

| Category | ASN100 | Placebo | Total |
|---|---|---|---|
| | (N=###) | (N=###) | (N=###) |
| | n (%) | n (%) | n (%) |
| Any Adverse Event (AE) | ### (###.#) | ### (###.#) | ### (###.#) |
| Any Treatment-Emergent Adverse Event (TEAE) | ### (###.#) | ### (###.#) | ### (###.#) |
| Mild TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Moderate TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Severe TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Drug-Related TEAEs [1] | ### (###.#) | ### (###.#) | ### (###.#) |
| Serious AEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Drug-Related Serious AEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Serious AEs Leading to Death | ### (###.#) | ### (###.#) | ### (###.#) |
| TEAEs Leading to Discontinuation of Study Drug | ### (###.#) | ### (###.#) | ### (###.#) |
| Serious TEAEs Leading to Discontinuation of Study Drug | ### (###.#) | ### (###.#) | ### (###.#) |

Percentage is calculated using the number of subjects in the column heading as the denominator.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

[1] Drug-Related is based on the Investigator's assessment.

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


Data Last Modified: MM/DD/YYYY HH:MM
Table 14.3.1.2
Subjects with Treatment-Emergent Adverse Events (TEAEs)

# Subjects with Treatment-Emergent Adverse Events (TEAEs) By System Organ Class and Preferred Term Safety Population

| System Organ Class | ASN100<br>(N=###) | Placebo<br>(N=###) | Total<br>(N=###) |
|---|---|---|---|
| Preferred Term | n (%) | n (%) | n (%) |
| Subjects with any TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| System Organ Class 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 3 | ### (###.#) | ### (###.#) | ### (###.#) |
| System Organ Class 2 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 3 | ### (###.#) | ### (###.#) | ### (###.#) |

Coding is based on MedDRA Version 19.1.

Percentage is calculated using the number of subjects in the column heading as the denominator.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

Subjects with multiple adverse events will be counted only once per system organ class and preferred term.

25OCTOBER2018 

The layouts of the following tables will be the same as Table 14.3.1.2:

Table 14.3.1.3

Subjects with Treatment-Emergent Serious Adverse Events (TESAEs)

By System Organ Class and Preferred Term

Safety Population

Table 14.3.1.4

Subjects with Drug-Related Treatment-Emergent Adverse Events By System Organ Class and Preferred Term  $\hbox{Safety Population}$ 

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.3.1.5

Subjects with Treatment-Emergent Adverse Events (TEAEs) By System Organ Class, Preferred Term and Maximum Severity Safety Population

| System Organ Class<br>Preferred Term<br>Maximum Grade | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) | Total<br>(N=###)<br>n (%) |
|---|---|---|---|
| Subjects with any TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Mild | ### (###.#) | ### (###.#) | ### (###.#) |
| Moderate | ### (###.#) | ### (###.#) | ### (###.#) |
| Severe | ### (###.#) | ### (###.#) | ### (###.#) |
| System Organ Class 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Mild | ### (###.#) | ### (###.#) | ### (###.#) |
| Moderate | ### (###.#) | ### (###.#) | ### (###.#) |
| Severe | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Mild | ### (###.#) | ### (###.#) | ### (###.#) |
| Moderate | ### (###.#) | ### (###.#) | ### (###.#) |
| Severe | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |


Percentage is calculated using the number of subjects in the column heading as the denominator.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

If the same TEAE (based on preferred term) is reported for the same patient more than once, the TEAE is counted only once for that preferred term and at the highest severity.

25OCTOBER2018  Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

#### Table 14.3.1.6

Subjects with Treatment-Emergent Adverse Events (TEAEs)
By System Organ Class, Preferred Term and Relationship to Study Drug
Safety Population

| System Organ Class Preferred Term Strongest Relationship | ASN100<br>(N=###)<br>n (%) | Placebo<br>(N=###)<br>n (%) | Total<br>(N=###)<br>n (%) |
|---|---|---|---|
| Subjects with any TEAEs | ### (###.#) | ### (###.#) | ### (###.#) |
| Not Related | ### (###.#) | ### (###.#) | ### (###.#) |
| Related | ### (###.#) | ### (###.#) | ### (###.#) |
| System Organ Class 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Not Related | ### (###.#) | ### (###.#) | ### (###.#) |
| Related | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 1 | ### (###.#) | ### (###.#) | ### (###.#) |
| Not Related | ### (###.#) | ### (###.#) | ### (###.#) |
| Related | ### (###.#) | ### (###.#) | ### (###.#) |
| Preferred Term 2 | ### (###.#) | ### (###.#) | ### (###.#) |


Percentage is calculated using the number of subjects in the column heading as the denominator.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

If the same TEAE (based on preferred term) is reported for the same patient more than once, the TEAE is counted only once for that preferred term and at the strongest relationship to study drug.

Drug-Related is based on the Investigator's assessment.

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Arsanis, Inc.

Arsanis, Inc.

Protocol Number: ASN100-201


Data Last Modified: MM/DD/YYYY HH:MM
Table 14.3.2.1
Listing of Serious Adverse Events
Safety Population

| Treatment<br>Subject | VT: Verbatim Term/<br>PT: Preferred Term/<br>SOC:System Organ Class | Start Date/Time/Day<br>Stop Date/Time/Day<br>Duration (days) | TEAE?/<br>Severity | Related to<br>Study Drug | Action Taken/<br>Other Action Taken/<br>Outcome |
|---|---|---|---|---|---|
| ASN100<br>###-###-### | VT: XXXXXXXXXX/ | YYYY-MM-DD/HH:MM/## | Yes/ | NOT RELATED | DOSE NOT CHANGED/ |
| пип ипп ппп | PT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Continuing | SEVERE | NOT KEDATED | MEDICATION REQUIRED/ NOT RECOVERED/NOT RESOLVED |
| ###-###-### | VT: XXXXXXXXXXX/<br>PT: XXXXXXXXXXXXXXX/<br>SOC:XXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>## | Yes/<br>XXXXXXX | RELATED | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXX |
| ###-###-### | VT: XXXXXXXXXXX/<br>PT: XXXXXXXXXXX/<br>SOC:XXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>## | Yes/<br>XXXXXXXX | XXXXXXXXX | XXXXXXXXXX/<br>XXXXXX/<br>XXXXXXXXX |
| Placebo | | | | | |


Day = Study day and is based on the first dose of study drug which is day 1.

Duration is calculated using stop date of adverse event - start date of adverse event + 1.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

25OCTOBER2018 

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Table 14.3.2.2 Listing of Adverse Events Leading to Discontinuation of Study Drug Safety Population

| Treatment<br>Subject | VT: Verbatim Term/<br>PT: Preferred Term/<br>SOC:System Organ Class | Start Date/Time/Day<br>Stop Date/Time/Day<br>Duration (days) | SAE?/<br>TEAE?/<br>Severity | Related to<br>Study Drug | Action Taken/<br>Other Action Taken/<br>Outcome |
|---|---|---|---|---|---|
| ASN100 | | | | | |
| ###-###-### | VT: XXXXXXXXXXX/ PT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>Continuing | Yes/<br>Yes/<br>SEVERE | NOT RELATED | DOSE NOT CHANGED/ MEDICATION REQUIRED/ NOT RECOVERED/NOT RESOLVED |
| ###-###-## | VT: XXXXXXXXXXX/<br>PT: XXXXXXXXXXXXXXX/<br>SOC:XXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>## | Yes/<br>Yes/<br>XXXXX | RELATED | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXX |
| ###-###-### | VT: XXXXXXXXXXX/<br>PT: XXXXXXXXXXX/<br>SOC:XXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>## | No/<br>XXX/<br>XXXXXX | XXXXXXXXX | XXXXXXXXXX/<br>XXXXXXX/<br>XXXXXXXXX |
| Dlagobo | | | | | |

Placebo


Day = Study day and is based on the first dose of study drug which is day 1.

Duration is calculated using stop date of adverse event - start date of adverse event + 1.

A treatment-emergent adverse events (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation of study drug administration.

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


## Table 14.3.3.1 Summary of Laboratory Chemistry Parameters Safety Population

| Parameter (unit)<br>Visit | | ASN100<br>(N=###) | | | Placebo<br>(N=###) | | | Total<br>(N=###) | |
|---|---|---|---|---|---|---|---|---|---|
| Statistics | Baseline | Post | Change | Baseline | Post | Change | Baseline | Post | Change |
| Parameter 1 (unit) | | | | | | | | | |
| Baseline [1]<br>n | ### | | | ### | | | ### | | |
| Mean | ##.## | | | ##.## | | | ##.## | | |
| SD | ##.### | | | ##.### | | | ##.### | | |
| Minimum | ##.# | | | ##.# | | | ##.# | | |
| Median | ##.## | | | ##.## | | | ##.## | | |
| Maximum | ##.# | | | ##.# | | | ##.# | | |
| Day 2 | | | | | | | | | |
| n [2] | ### | ### | ### | ### | ### | ### | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| SD | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.### |
| Minimum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Day 4 | | | | | | | | | |
| n [2] | ### | ### | ### | ### | ### | ### | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| SD | ##.### | ##.### | ##.## | ##.## | ##.## | ##.## | ##.### | ##.## | |
| Minimum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |

<< Programming note: Repeat for all scheduled visits. Parameters to be included: Alanine aminotransferase (ALT), Albumin, Alkaline phosphatase, Aspartate aminotransferase (AST), Bicarbonate, Blood urea nitrogen, Calcium, Chloride, Creatinine, Direct bilirubin, Glucose, Phosphorus, Potassium, Sodium, Total bilirubin, and Total protein>>

25OCTOBER2018 

<sup>[1]</sup> Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

<sup>[2]</sup> n is the number of subjects with both baseline and post-baseline measurements.

The layouts of the following tables will be the same as Table 14.3.3.1:

Table 14.3.3.2

Summary of Laboratory Hematology Parameters

Safety Population

<< Parameters to be included: Absolute neutrophil count, Hematocrit, Hemoglobin, Platelet count, Red blood cell (RBC) count, White blood cell (WBC) count with differential (basophils, eosinophils, lymphocytes, monocytes, and neutrophils), RBC indices mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), and "Reticulocytes.">>>

Table 14.3.3.3
Summary of Laboratory Coagulation Parameters
Safety Population

<< Parameters to be included: Prothrombin time and Partial thromboplastin time (PTT)>>

Table 14.3.3.4
Summary of Laboratory Urinalysis Parameters
Safety Population
<< Parameters to be included: pH and Specific Gravity>>

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc. Protocol No. ASN100-201

Arsanis, Inc.

Protocol Number: ASN100-201


Sì

| | | Tabl | e 14.3.3.5 | |
|------|-------|------|--------------|------------|
| hift | Table | for | Hematology | Parameters |
| | Sa | fets | , Population | n |

| Parameter (unit) | | I | Low | N | ormal | F | ligh | Mi | ssing | I | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Baseline [1] | n | (응) | n | (%) | n | (%) | n | (%) | n | (%) |
| Parameter 1 (unit) | | | | | | | | | | | |
| | | | 7 H H H H H N | 0.0.0 | ( 11 11 11 11 ) | шшш | (###.#) | шшш | (###.#) | 11 11 11 | (###.#) |
| ASN100 (N=###) | Low | ### | (###.#) | ### | (###.#) | ### | (###•#) | ### | (###•#) | ### | (###•#) |
| ASN100 (N=###) | Low<br>Normal | | (###.#) | | (###.#) | | (###.#) | | (###.#) | | (###.#) |
| ASN100 (N=###) | | ### | | ### | | ### | | ### | | ### | |
| ASN100 (N=###) | Normal | ### | (###.#) | ###<br>### | (###.#) | ###<br>### | (###.#) | ###<br>### | (###.#) | ###<br>### | (###.#) |

Placebo (N=###)

<< Programming note: Parameters to be included: Hematocrit, Hemoglobin, Platelets, White blood cell count and differential including Basophils, Neutrophils, Lymphocytes, Monocytes, and Eosinophils>>

[1] Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

25OCTOBER2018  Protocol No. ASN100-201

Arsanis, Inc.

Protocol Number: ASN100-201


#### Table 14.3.3.6 Shift Table for Chemistry Parameters Safety Population

Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

| Parameter (unit) | | | <lln< th=""><th></th><th>Normal</th><th></th><th>JLN and<br/>=3xULN</th><th></th><th>xULN and<br/>=5xULN</th><th>&gt;</th><th>5xULN</th><th>М</th><th>issing</th><th></th><th>Total</th></lln<> | | Normal | | JLN and<br>=3xULN | | xULN and<br>=5xULN | > | 5xULN | М | issing | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Baseline [1] | n | (왕) | n | (왕) | n | (왕) | n | (왕) | n | (왕) | n | (왕) | n | (왕) |
| Parameter 1 (unit) | | | | | | | | | | | | | | | |
| ASN100 (N=###) | <lln< td=""><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td><td>###</td><td>(###.#)</td></lln<> | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | Normal | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | >ULN and $<=3xULN$ | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | >3xULN and $<=5xULN$ | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | >5xULN | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | Missing | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |
| | Total | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) | ### | (###.#) |

<< Programming note: Parameters to be included: ALT, AST, Total Bilirubin, Creatinine, and ALP>>

25OCTOBER2018 

<sup>[1]</sup> Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

Arsanis, Inc.
Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Table 14.3.3.7

Number (%) of Subjects with Prespecified Potentially Clinically Significant Abnormal Post-Baseline Liver Function Tests
Safety Population

| Parameter<br>Category | ASN100<br>(N=###)<br>n/N' (%) | Placebo<br>(N=###)<br>n/N' (%) | Total<br>(N=###)<br>n/N' (%) |
|---|---|---|---|
| Subjects with a valid post-baseline value, N' | ### | ### | ### |
| ALT | | | |
| >=3xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| >=5xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| AST | | | |
| >=3xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| >=5xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| ALT or AST | | | |
| >=3xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| >=5xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |

 $\hbox{Percentage is calculated using $\tt N'$, the number of subjects with a valid post-baseline assessment as the denominator. } \\$ 

25OCTOBER2018 

<sup>\*</sup> Potential Hy's Law case is defined as ALT or AST >=3xULN, Total bilirubin >=2xULN and ALP <= 2xULN.

Arsanis, Inc.
Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Table 14.3.3.7

Number (%) of Subjects with Prespecified Potentially Clinically Significant Abnormal Post-Baseline Liver Function Tests
Safety Population

| Parameter<br>Category | ASN100<br>(N=###)<br>n/N' (%) | Placebo<br>(N=###)<br>n/N' (%) | Total<br>(N=###)<br>n/N' (%) |
|---|---|---|---|
| Total bilirubin | | | |
| >=1.5xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| >=2xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| ALP | | | |
| >=1.5xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| >=3xULN | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| ALT or AST $>=3xULN$ and Total bilirubin $>=2xULN$ | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |
| Potential Hy's Law case * | ###/### (##.#) | ###/### (##.#) | ###/### (##.#) |

Percentage is calculated using N', the number of subjects with a valid post-baseline assessment as the denominator.

25OCTOBER2018 

<sup>\*</sup> Potential Hy's Law case is defined as ALT or AST >=3xULN, Total bilirubin >=2xULN and ALP <= 2xULN.

Arsanis, Inc.

Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Protocol Number: ASN100-201 Page 1 of # Data Last Modified: MM/DD/YYYY HH:MM

Table 14.3.3.8

Listing of Subjects with Prespecified Potentially Clinically Significant Abnormal Post-Baseline Liver Function Findings Safety Population

| Treatment<br>Subject | Parameter | (Unit) | Normal Range | Visit | Date and Time<br>of Collection/Day | Result | Met Criteria |
|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | xxxxxxx | (XXXX) | ##.#-##.# | Day 1 Pre-dose<br>XXXXXXXXX<br>XXXXXXXX<br>XXXXXXXXX | YYYY-MM-DD/HH:MM/## YYYY-MM-DD/HH:MM/## YYYY-MM-DD/HH:MM/## YYYY-MM-DD/HH:MM/## | ## | ALT >= 3xULN |
| | xxxxxxx | (XXXX) | ##.#-##.# | Day 1 Pre-dose<br>XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | ##.#<br>##.#<br>##.# | AST >= 3xULN |
| ###-###-### | xxxxxxx | (XXXX) | ##.#-##.# | Day 1 Pre-dose<br>XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | ##.#<br>##.#<br>##.# | ALP >= 1.5xULN |
| Placebo | | | | | | | |

Day = Study day and is based on the first dose of study drug which is day 1.

25OCTOBER2018 

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Arsanis, Inc.

Protocol Number: ASN100-201


Table 14.3.4
Summary of Vital Signs
Safety Population

| Parameter (unit)<br>Visit<br>Statistics | Baseline | ASN100<br>(N=###)<br>Post | Change | Baseline | Placebo<br>(N=###)<br>Post | Change | Baseline | Total<br>(N=###)<br>Post | Change |
|---|---|---|---|---|---|---|---|---|---|
| Parameter 1 (unit) | | | | | | | | | |
| Baseline [1]<br>n | ### | | | ### | | | ### | | |
| Mean | ##.## | | | ##.## | | | ##.## | | |
| SD | ##.### | | | ##.### | | | ##.### | | |
| Minimum | ##.# | | | ##.# | | | ##.# | | |
| Median | ##.## | | | ##.## | | | ##.## | | |
| Maximum | ##.# | | | ##.# | | | ##.# | | |
| Day 1 | | | | | | | | | |
| n [2] | ### | ### | ### | ### | ### | ### | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| SD | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.### |
| Minimum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Day 2 | | | | | | | | | |
| n [2] | ### | ### | ### | ### | ### | ### | ### | ### | ### |
| Mean | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| SD | ##.## | ##.## | ##.### | ##.### | ##.## | ##.## | ##.## | ##.### | ##.## |
| Minimum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |
| Median | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## | ##.## |
| Maximum | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# | ##.# |

<< Program note: Repeat for all scheduled visits; Parameters also to be included: Systolic BP (mmHg), Diastolic Blood Pressure (mmHg), Pulse (bpm), Respiratory Rate (rpm), Temperature (C), pH, PaO2 (mmHg), PaCO2 (mmHg), and SpO2 (%)>>

25OCTOBER2018 

<sup>[1]</sup> Baseline is defined as the last measurement or assessment prior to the first and only dose of study drug.

<sup>[2]</sup> n is the number of subjects with both baseline and post-baseline measurements.

### Figure Mock-Ups

| FIGURE 14.2.1.1 |
|---|
| Kaplan-Meier Plot of Overall Survival (Days) by Treatment |
| Modified Intent-to-Treat Population |
| FIGURE 14.2.2.1 |
| Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22<br>Based on Sponsor-Defined Outcome (SDO1) |
| Modified Intent-to-Treat Population |
| FIGURE 14.2.2.2 |
| Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22<br>Based on Sponsor-Defined Outcome (SDO2) |
| Modified Intent-to-Treat Population |
| FIGURE 14.2.2.3 |
| Additional Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO1) |
| Modified Intent-to-Treat Population |
| FIGURE 14.2.2.4 |
| Additional Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO2) |
| Modified Intent-to-Treat Population |
| FIGURE 14.2.2.5 |
| Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 |
| Determined by Investigator's Judgement and Review Meeting's Determination of S. aureus as a Causative Pneumonia Pathogen |
| Modified Intent-to-Treat Population |

25OCTOBER2018 

Arsanis, Inc.
Protocol Number: ASN100-201

Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Figure 14.2.1.1
Kaplan-Meier Plot of Overall Survival (Days) by Treatment
Modified Intent-to-Treat Population



25OCTOBER2018 

CONFIDENTIAL

Arsanis, Inc. Protocol Number: ASN100-201

Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Page 1 of # Data Last Modified: MM/DD/YYYY HH:MM

Figure 14.2.2.1 Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO1) Modified Intent-to-Treat Population



Note: Subjects who did not develop S. aureus pneumonia, discontinued from the study, or died prior to Day 22 will be considered censored.

25OCTOBER2018 

#### The layouts of the following tables will be the same as Figure 14.2.2.1:

Figure 14.2.2.2

Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO2)

Modified Intent-to-Treat Population

<< Programming note: For figures 14.2.2.3 and 14.2.2.4, footnote will use "Note: Discontinuation from the study due to any cause up to but not including Day 22 will be considered as an event.">>

Figure 14.2.2.3

Additional Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO1)

Modified Intent-to-Treat Population

Figure 14.2.2.4

Additional Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22 Based on Sponsor-Defined Outcome (SDO2)

Modified Intent-to-Treat Population

<< Programming note: For figure 14.2.2.5, no footnote will be used>>

Figure 14.2.2.5

Kaplan-Meier Plot of Time to S. aureus Pneumonias Up to But Not Including Day 22

Determined by Investigator's Judgement and Review Meeting's Determination of S. aureus as a Causative Pneumonia Pathogen

Modified Intent-to-Treat Population

25OCTOBER2018 

### **Listings Mock-ups**

| LISTING 16.2.1.1 | 107 |
|-------------------------------------------------|-----|
| Screen Failures | |
| All Subjects | |
| LISTING 16.2.1.2 | 108 |
| Subject Disposition | |
| Intent-to-Treat Population | |
| LISTING 16.2.1.3 | 109 |
| Subject Randomization | |
| All Subjects | |
| LISTING 16.2.1.4 | 110 |
| Sub-Study for Subjects Diagnosed with Pneumonia | |
| All Subjects | |
| LISTING 16.2.2 | 111 |
| Protocol Deviations | |
| Intent-to-Treat Population | |
| LISTING 16.2.3.1 | 112 |
| Subject Population | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.1 | 113 |
| Demographics | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.2 | 114 |
| Smoking Medical History | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.3 | 115 |
| Medical History | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.4 | 116 |
| Prior and Concomitant Medications | |
| Intent-to-Treat Population | |

| LISTING 16.2.4.5 | 117 |
|----------------------------------------------------|-----|
| Concomitant Procedure and Non-Drug Therapies | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.6 | 118 |
| Ventilator Status | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.7 | 119 |
| Risk Factors for Ventilator - Associated Pneumonia | |
| Intent-to-Treat Population | |
| LISTING 16.2.4.8 | 120 |
| VAP Prevention | |
| Intent-to-Treat Population | |
| LISTING 16.2.5.1 | 121 |
| Study Drug Administration | |
| Intent-to-Treat Population | |
| LISTING 16.2.5.2 | 122 |
| Pharmacokinetic Serum Sampling | |
| Intent-to-Treat Population | |
| LISTING 16.2.5.3 | 123 |
| Pharmacokinetic BAL Sampling | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.1 | 124 |
| ETA Specimen Culture | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.2 | 125 |
| Respiratory Culture from Local Laboratory | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.3 | 126 |
| Blood Culture from Local Laboratory | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.4 | 127 |
| Other Cultures from Local Laboratory | |
| Intent-to-Treat Population | |

| LISTING 16.2.6.5 | 128 |
|-------------------------------------------------------|-----|
| Nasal Swab Specimen | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.6 | 129 |
| Microbiological Results from Central Laboratory | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.7 | 130 |
| Radiograph and Imaging | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.8 | 131 |
| Clinical Signs and Symptoms - Pneumonia | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.9 | 132 |
| Clinical Signs and Symptoms and Pneumonia Progression | |
| Pilot Rx Arm Amendment | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.10 | 133 |
| Investigator Clinical Outcome of Pneumonia | |
| Pilot Rx Arm Amendment | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.11 | 134 |
| Hospitalization Course and Discharge | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.12 | 135 |
| Anti-Drug Antibodies Sample Collection | |
| Intent-to-Treat Population | |
| LISTING 16.2.6.13 | 136 |
| Survival Status | |
| Intent-to-Treat Population | |
| LISTING 16.2.7.1 | 137 |
| Adverse Events | |
| Intent-to-Treat Population | |

| LISTING 16.2.7.2 | 138 |
|-----------------------------------------------|-----|
| Serious Adverse Events | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.1 | 139 |
| Central Laboratory Parameters - Chemistry | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.2 | 140 |
| Central Laboratory Parameters - Hematology | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.3 | 140 |
| Central Laboratory Parameters - Urinalysis | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.4 | 140 |
| Central Laboratory Parameters - Coagulation | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.5 | 140 |
| Central Laboratory Parameters - Procalcitonin | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.6 | 141 |
| Urine Pregnancy Test from Local Laboratory | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.7 | 142 |
| Vital Signs | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.8 | 143 |
| 12-Lead Electrocardiogram | |
| Intent-to-Treat Population | |
| LISTING 16.2.8.9 | 144 |
| Physical Examination | |
| Intent-to-Treat Population | |

Arsanis, Inc.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

Listing 16.2.1.1 Screen Failures All Subjects

| e of Screen Failure 1 | Reason for Screen Failure |
|-----------------------|-----------------------------------------|
| YY-MM-DD | ××××××××××××××××××××××××××××××××××××××× |
| Y-MM-DD | XXXXXXXXXXXXXXXXXXXXX |
| Y-MM-DD ( | Other: XXXXXXXXXXXXXX |
| Y-MM-DD | xxxxxxxxx |
| YY-MM-DD | XXXXXXXXXXXXXXXXXXXX |
| 7 | Y-MM-DD<br>Y-MM-DD<br>Y-MM-DD |

Note: A subject was considered a screen failure if they were enrolled in the trial and underwent daily screening of endotracheal aspirates for the presence of S. aureus.

Arsanis, Inc.

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

## Listing 16.2.1.2 Subject Disposition Intent-to-Treat Population

| Treatment<br>Subject | Complete Study?/<br>Reason Study<br>Not Completed [1] | Date/Study Day of Completion<br>or Early Termination [2] | Prematurely Unblinded? |
|---|---|---|---|
| ASN100<br>###-###-###<br>###-###-###<br>###-### | No/XXXXXXXXXXXXXXX<br>No/Other:XXXXXXXXX<br>Yes | YYYY-MM-DD/##<br>YYYY-MM-DD/##<br>YYYY-MM-DD/## | No<br>Yes<br>No |
| Placebo | | | |

Day = Study day and is based on first dose of study drug which is Day 1.

<sup>[1]</sup> Study considered complete if subject completed the study through the Day 90 Safety Visit.

<sup>[2]</sup> If a subject completed the study, date of completion is displayed. Otherwise, date of early termination is displayed.
Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.1.3 Subject Randomization All Subjects

| Treatment<br>Subject | Protocol<br>Version | Met All Inclusion and<br>No Exclusion Criteria?/<br>Criteria Not Satisfied | Heavily<br>Colonized<br>with<br>S. aureus? | Remain<br>Mechanically<br>Ventilated?* | Probable<br>Survival?** | Date/Time of<br>Randomization | Kit ID | Receiving<br>Antibiotic? [1] |
|---|---|---|---|---|---|---|---|---|
| | 02May2017 | Yes<br>No/INCL##, EXCL## | Yes<br>Yes | Yes<br>No | Yes | YYYY-MM-DD/HH:MM<br>YYYY-MM-DD/HH:MM | | Yes<br>No |

#### Placebo

#### Screen Failure

<sup>\*</sup> In investigator's opinion, subject will require ongoing ventilator support for at least 48 hrs.

<sup>\*\*</sup> In Investigator's opinion, survival beyond 72 hrs post-randomization is expected.

<sup>[1]</sup> Is the subject receiving concomitant anti-staphylococcal antibiotics at the time of randomization that are potentially active against S. aureus pneumonia?

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.1.4 Sub-Study for Subjects Diagnosed with Pneumonia All Subjects

| Treatment<br>Subject | Presumed S.aureus Pneumonia at Randomization? | Previous and/or Current Anti-staphylococcal<br>Antibiotic Exposure* |
|---|---|---|
| ASN100 | | |
| ###-##-## | Yes | <24 hours |
| ###-###-## | Yes | >= 24 hours |
| ###-###-## | No | < 72 hours |
| ###-###-## | Yes | >= 72 hours |
| ###-###-## | XXX | ########### |
| Placebo | | |
| Screen Failure | | |

<sup>\*</sup> Previous and/or current anti-staphylococcal antibiotic exposure that is potentially effective against S. aureus pneumonia.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.2 Protocol Deviations Intent-to-Treat Population

| Treatment<br>Subject | Occurrence<br>Date/Day | Deviation<br>Type | Protocol Deviation | Action | CSR<br>Reportable? |
|---|---|---|---|---|---|
| ASN100<br>###-###-### | YYYY-MM-DD/## | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No<br>XXX |
| ###-###-### | YYYY-MM-DD/## | XXXXXXXX | xxxxxxxxxxxxxxxxx | xxxxxxxxxxx xxx | |
| ###-###-### | YYYY-MM-DD/## | XXXXXXXXXXX<br>XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| ###-###-### | YYYY-MM-DD/## | xxxxxxxxx xxxxxx | xxxxxxxxxxxxx | xxxxxxxxxxxx xxx | |
| Placebo | | | | | |

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

## Listing 16.2.3.1 Subject Population Intent-to-Treat Population

| No<br>Yes |
|-----------|
| Yes |
| Yes |
| Yes |
| Yes |
| Yes |

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.4.1 Demographics Intent-to-Treat Population

| Treatment<br>Subject | Date of<br>Informed Consent | Protocol<br>Version | Date of<br>Birth | Age at Enrollment (Years) | Sex | Ethnicity [1] | Race |
|---|---|---|---|---|---|---|---|
| ASN100 | | | | | | | |
| ###-##-## | YYYY-MM-DD | 02MAY2017 | YYYY-MM | ## | F | HT | XXXXXXX |
| ###-##-### | YYYY-MM-DD | 16NOV2016 | YYYY-MM | ## | M | NHT | Other: XXXXXXXX |
| ###-##-## | YYYY-MM-DD | DDMMMYYYY | MM-YYYY | ## | M | NR | XXXXXXX |
| ###-##-### | YYYY-MM-DD | DDMMMYYYY | MM-YYYY | ## | M | UNK | XXXXXXX |
| ###-##-### | YYYY-MM-DD | DDMMMYYYY | MM-YYYY | ## | F | NHT | XXXXXXX |
| ###-##-## | YYYY-MM-DD | DDMMMYYYY | YYYY-MM | ## | M | NHT | XXXXXXX |

<sup>[1]</sup> Ethnicity: HT = Hispanic or Latino, NHT = Not Hispanic or Latino, NR = Not Reported, UNK = Unknown.

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.4.2 Smoking Medical History Intent-to-Treat Population

| Treatment<br>Subject | History of Smoking? | Packs Smoked<br>Per Week | Duration of<br>Smoking (Years) |
|---|---|---|---|
| ASN100<br>###-###-###<br>###-###-###<br>###-### | Never<br>Current<br>Former | # | ##<br>## |
| Placebo | | | |

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.4.3 Medical History Intent-to-Treat Population

| Treatment<br>Subject | Event/<br>Diagnosis | Start Date/Day | End Date/Day |
|---|---|---|---|
| ASN100<br>###-###-### | xxxxxxxxxxx<br>xxxxx<br>xxxxxxxxxxxxxxxxxxxx | YYYY-MM-DD/##<br>YYYY-MM-DD/## | YYYY-MM-DD/##<br>Ongoing<br>YYYY-MM-DD/## |
| ###-###-### | XXXXXXXXXX | YYYY-MM-DD/## | YYYY-MM-DD/## |
| Placebo | | | |

Day = Study day and is based on first dose of study drug which is Day 1.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.4.4 Prior and Concomitant Medications Intent-to-Treat Population

| Treatment<br>Subject | VT: Medication Name<br>PT: Preferred Term<br>ATC:Medication Class | Indication | Dose/<br>Unit | Frequency/<br>Route | Start Date/Time/Day/<br>Stop Date/Time/Day |
|---|---|---|---|---|---|
| ASN100<br>###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx | YXXXXXXXXX/<br>YXXXXXXXX | xxxxxxxx/<br>xxxxxxxxx | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/## |
| ###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXXXX/<br>Other: XXXXX | Other: XXX/<br>Other: XXXX | YYYY-MM-DD/HH:MM/##<br>Ongoing |

Placebo

Coding is based on WHO Drug Dictionary Sept 2016E B2.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.4.5 Concomitant Procedure and Non-Drug Therapies Intent-to-Treat Population

| Treatment<br>Subject | VT: Procedure/Non-Drug Therapy<br>PT: Preferred Term<br>SOC:System Organ Class | Indication | Start Date/Time/Day<br>Stop Date/Time/Day |
|---|---|---|---|
| ASN100 | | | |
| ###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## |
| | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## |
| ###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx | YYYY-MM-DD/HH:MM/##<br>Ongoing |
| Placebo | | | |


Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.4.6 Ventilator Status Intent-to-Treat Population

| Treatment<br>Subject | Underlying<br>Condition<br>[1] | Start Date/Time of<br>Initial Intubation | Visit | Mechanically<br>Ventilated at<br>This Visit? | Type [2] | FiO2: | * PEEP**<br>(cm H2O) | Is Subject Currently<br>Extubated or Since<br>Previous Assessment? | Date/Time of Extubation |
|---|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | T, CI, NI | YYYY-MM-DD/HH:MM | XXXXX<br>XXXXX<br>XXXXX | Yes<br>No<br>Yes | E<br>T | ## | ##### | Yes<br>Yes<br>No | YYYY-MM-DD/HH:MM<br>YYYY-MM-DD/HH:MM |
| ###-###-### | Other: XXXXX | X YYYY-MM-DD/HH:MM | XXXXX<br>XXXXX<br>XXXXX | Yes<br>No<br>Yes | OTH<br>E | ## | ##### | Yes<br>Yes<br>No | YYYY-MM-DD/HH:MM<br>YYYY-MM-DD/HH:MM |

Placebo

[1] T = Trauma, CI = Cardiovascular Impairment, NI = Neurological Impairment, PI = Pulmonary Impairment, Other.

<sup>[2]</sup> E = Endotracheal, T = Tracheotomy, OTH = Other.

<sup>\*</sup> Predominant FiO2 setting (%) in the past 24 hours.

<sup>\*\*</sup> Predominant PEEP setting (cm H2O) in the past 24 hours.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.4.7 Risk Factors for Ventilator - Associated Pneumonia Intent-to-Treat Population

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.4.8 VAP Prevention Intent-to-Treat Population

| Treatment Subject | Visit | VAP<br>Prevention? | Techniques Applied | Silver Impregnated<br>Endotracheal Tube Used? |
|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | Yes | Elevation of head of the bed; Daily sedation vacations and assessment of readiness to extubate; Peptic ulcer disease prophylaxis; Deep vein thrombosis prophylaxis; Daily oral care with chlorhexidine or equivalent; | No |
| ###-###-### | XXXXXX | No | | Unknown |
| ###-###-### | XXXXXX | Yes | Elevation of head of the bed; Peptic ulcer disease prophylaxis; | Yes |
| ###-###-### | XXXXXX | No | | Yes |

Placebo

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.5.1 Study Drug Administration Intent-to-Treat Population

| Treatment<br>Subject | Date/Time/Day of<br>Drug Preparation | Bag | Infusion<br>Start Date/Time/Day/<br>End Date/Time/Day | Total Volume<br>Infused (mL)/<br>Entire Bag<br>Infused? | Line Flushed?/<br>Reason Not Done | True Stop Time of Flush Known?/<br>Est. Stop Time of Flush Aval.?*/<br>Stop Time |
|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | YYYY-MM-DD/HH:MM/## | А | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/## | #####/<br>Yes | Yes | Yes/-/HH:MM |
| | | В | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/## | #####/<br>No | No/XXXXXXX | |
| ###-###-### | YYYY-MM-DD/HH:MM/## | А | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/## | #####/<br>Yes | Yes | No/Yes/HH:MM |
| | | В | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/## | #####/<br>Yes | Yes | No/No/ |

#### Placebo

<sup>\*</sup> Only collected if line was flushed and if the true stop time of flush not known.

Protocol Number: ASN100-201


Listing 16.2.5.2
Pharmacokinetic Serum Sampling

Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Intent-to-Treat Population

Date/Time/Day of Collection/
Subject Visit Time Point Not performed - Reason Not Done

ASN100
###-###-### Day 1 +15 min YYYY-MM-DD/HH:MM/##

6 hrs Site Error Other: XXXXXXXX Day 2 +/- 1 hr relative to BAL fluid collection YYYY-MM-DD/HH:MM/## +/- 1 hr relative to BAL fluid collection YYYY-MM-DD/HH:MM/## Day 3 Day 4 YYYY-MM-DD/HH:MM/## Day 7 YYYY-MM-DD/HH:MM/## Day 14 YYYY-MM-DD/HH:MM/## Day 22 YYYY-MM-DD/HH:MM/##

Placebo

Day = Study day and is based on first dose of study drug which is Day 1.

122

Protocol Number: ASN100-201


Placebo

Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.5.3 Pharmacokinetic BAL Sampling Intent-to-Treat Population

| Treatment | Visit | Collected?/ | Collection |
|-------------|-------|---------------------|---------------------|
| Subject | | Reason Not Done | Date/Time/Day |
| ASN100 | Day 2 | Yes | YYYY-MM-DD/HH:MM/## |
| ###-###-### | Day 3 | No/Other: XXXXXXXXX | |

Day = Study day and is based on first dose of study drug which is Day 1.

123

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

#### Listing 16.2.6.1 ETA Specimen Culture Intent-to-Treat Population

| Treatment<br>Subject | Visit | ETA Collected?/<br>Reason Not Done | Date/Time/Day<br>of Collection | Identified?<br>Number of<br>Unique<br>Organisms | /<br>Genus and Species | MRSA or<br>MSSA? [1] | Result | Isolate<br>Stored for<br>Shipment?/<br>Local Lab ID |
|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | Yes | YYYY-MM-DD/HH:MM/## | Yes/3 | Staphylococcus aureus<br>XXXXXXXXXXXXXXXXX<br>Other: XXXXXXXXXX | MRSA | 1+<br>>10^5<br>3+ | Yes/###<br>No<br>No |
| ###-###-### | XXXXXX | Yes | YYYY-MM-DD/HH:MM/## | No | | | | |
| ###-###-## | XXXXXX | No/Other: XXXXXXX | | | | | | |

#### Placebo

<sup>[1]</sup> MRSA or MSSA: MRSA, MSSA, or ND = Not Determined. Collected only if Staphylococcus aureus specified.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.6.2 Respiratory Culture from Local Laboratory Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day<br>Sample Collected<br>or Reason Not Done | Type[1]/<br>Squ.[2]/<br>PMNs[3] | Pathogen<br>Isolated?/<br>Number of<br>Unique<br>Pathogens | Semi-quantitative<br>or Quantitative?/<br>Specify Pathogen | MRSA or<br>MSSA? [4] | Result | Stored for<br>Shipment?/<br>Local Lab ID |
|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | YYYY-MM-DD/HH:MM/<br>## | XXXX/<br>Yes/<br>No | Yes/3 | Quantitative/<br>Staphyloccus<br>aureus | MRSA | >##x10^6 | Yes/### |
| | | | | | Semi-quantitative/<br>Escherichia coli | | #+ | Yes/#### |
| | | | | | XXXXXXX/<br>Other:XXXXXXXXXXXX | | ## | No |
| | xxxxxx | YYYY-MM-DD/HH:MM/<br>## | Oth:XXXXX<br>XXXXXXX/<br>Yes/<br>Yes | No | | | | |
| ###-###-## | XXXXXXX | No/Subject Refused | | | | | | |
| | XXXXXXX | No/Other: XXXXXXX | | | | | | |
| Placebo | | | | | | | | |

<sup>[1]</sup> NBB = Non-Bronchoscopic BAL, PBS = Protected brush specimen, ES = Expectoracted or induced sputum, Oth = Other.

<sup>[2]</sup> Did the specimen contain <10 squamous epithelial cells/100 x field? Collected if type is expectorated or induced sputum.

<sup>[3]</sup> Did the specimen contain >25 PMNs/100 x field? Collected if type is expectorated or induced sputum.

<sup>[4]</sup> MRSA or MSSA: MRSA, MSSA, or ND = Not Determined. Collected ony if Staphylococcus aureus specified.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.6.3 Blood Culture from Local Laboratory Intent-to-Treat Population

| Treatment<br>Subject | Visit | Collected?/<br>Reason Not Done | Date/Time/Day<br>of Collection | Pathogen<br>Isolated?/<br>Number of<br>Unique | Genus and Species | MRSA or<br>MSSA? [1] | Stored for<br>Shipment?/<br>Local Lab ID |
|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | Yes | YYYY-MM-DD/HH:MM/## | Yes/2 | Staphylococcus aureus<br>Other: XXXXXXXXXXXXXXXXX<br>Enterococcus faecium | MRSA | No |
| | XXXXXXX | Yes | YYYY-MM-DD/HH:MM/## | Yes/1 | xxxxxxxxxxxxxxxxxx | | |

###-###-## XXXXXXX No/Other: XXXXX

#### Placebo

Day = Study day and is based on first dose of study drug which is Day 1.

[1] MRSA or MSSA: MRSA, MSSA, or ND = Not Determined. Collected ony if Staphylococcus aureus specified.

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.6.4 Other Cultures from Local Laboratory Intent-to-Treat Population

| Treatment<br>Subject | Visit | Other<br>Specimen<br>Collected?/<br>Reason Not Done | S. aureus<br>Isolated? | Source | Date/Time/Day<br>of Collection | Number of<br>Unique<br>S. aureus | MRSA or<br>MSSA? [1] | Isolate Stored<br>for Shipment to<br>Central Lab | Local<br>Lab<br>ID |
|---|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | Yes | Yes | Urine<br>XXXXXX<br>Other:XXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | 2<br>0<br>1 | MRSA<br>MRSA | Yes<br>No<br>Yes | #### |
| | XXXXXXX | Yes | No | | | | | | |
| ###-###-### | XXXXXXx | No/Other: XXX | | | | | | | |
| Placebo | | | | | | | | | |

Day = Study day and is based on first dose of study drug which is Day 1. [1] MRSA or MSSA: MRSA, MSSA, or ND = Not Determined.

Program Name: XXXX.sas Protocol Number: ASN100-201 Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM


Listing 16.2.6.5 Nasal Swab Specimen Intent-to-Treat Population

| Treatment<br>Subject | Swab Collected from Right Nostril? | Date/Time/Day of Right<br>Nostril Collection | Swab Collected from Left Nostril? | Date/Time/Day of Left<br>Nostril Collection | Reason Not<br>Collected* |
|---|---|---|---|---|---|
| ASN100<br>###-###-### | Yes | YYYY-MM-DD/HH:MM/## | No | | xxxxxxxxxxxx |
| ###-###-##<br>###-###-### | Yes<br>Yes | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | Yes<br>Yes | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | |
| ###-###-## | No | IIII-MM-DD/nn:MM/## | No | IIII-MM-DD/nn:MM/## | XXXXXXXXXXXXX |

Placebo

Day = Study day and is based on first dose of study drug which is Day 1.

128

<sup>\*</sup> Applies to swab collection from either right or left nostril.

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.6.6 Microbiological Results from Central Laboratory Intent-to-Treat Population

| Treatment<br>Subject | Visit | Specimen Collection<br>Date/Time/Day | Source of | Local<br>Specimen<br>Number | Central<br>Genus and Species | Inducible<br>Clindamycin<br>Resistance | Antimicrobial | MIC(1<br>Result | ug/mL)<br>Interp. |
|---|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXXX | YYYY-MM-DD/HH:MM/## | ETA | #### | Staphylococcus aureus | s Negative | Ampicillin<br>Ceftaroline<br>XXXXXXXXX<br>XXXXXXXXX | 0.120<br>20.000<br>##.###<br><##### | S<br>I<br>R<br>NA |
| | XXXXXX | YYYY-MM-DD/HH:MM/## | Respiratory | #### | Klebsiella pneumoniae | e Positive | XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX | ##.##<br>##.##<br>##.##<br>##.## | I<br>I<br>R<br>I |
| | | | NASAL SWAB | #### | Staphylococcus aureus | s Negative | XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX | ##.##<br>##.##<br>##.##<br>##.## | I<br>I<br>NA<br>I |

Placebo

Day = Study day and is based on first dose of study drug which is Day 1. MIC Interpretation: S = Susceptible, I = Intermediate, R = Resistant, NA = Not Available.

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

#### Listing 16.2.6.7 Radiograph and Imaging Intent-to-Treat Population

| Treatment<br>Subject | Visit | Imaging Preformed?/<br>Reason Not Done | Туре | Date/Time/Day<br>Performed | Infiltrates Present?/<br>Consistent with<br>Pneumonia? | Description of<br>Infiltrates |
|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | XXXXX | Yes<br>Yes | XXXXXXX<br>Other: XXXXXXXX | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | Yes/Yes<br>No | Other: XXXXXXX |
| ###-###-### | XXXXX<br>XXXXX<br>XXXXX | No/Other: XXXXX No/XXXXXXXXXXXXX Yes | xxxxxxxx | YYYY-MM-DD/HH:MM/## | Yes/No | ***** |

#### Placebo

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.6.8 Clinical Signs and Symptoms - Pneumonia Intent-to-Treat Population

| Treatment<br>Subject | Visit | Item | Result |
|---|---|---|---|
| ASN100 | | | |
| ###-##-## | XXXXXX | Was a chest assessment performed?/Reason if not assessed | Yes |
| | | Date/Time/Day performed | YYYY-MM-DD/HH:MM/## |
| | | Does chest x-ray show new or progressive infiltrates suggestive of pneumonia? | No |
| | | Has the subject been hospitalized for > 48 hours? | Yes |
| | | Has the subject received mechanical ventilation via an | |
| | | endotracheal or nasotracheal tube for >= 48 hours? | Yes |
| | | Has the subject developed clinical signs and symptoms within 7 days | |
| | | following hospital discharge? | No |
| | | Has the subject developed new onset or worsening pulmonary signs or symptoms | |
| | | or the requirement for mechanical ventilation? | No |
| | | Was there a need for acute changes in ventilator support to enhance oxygenation | |
| | | or to the amount of PEEP? | No |
| | | Was there new onset of suctioned respiratory secretions? | No |
| | | Was temperature > 38°C or < 35°C? No | |
| | | Was WBC count >= 10,000 cel1/mm3 or <= 4500 cel1/mm3? | No |
| | | Was > 15% immature neutrophils (bands) seen on peripheral blood smear? | No |
| | | Was diagnosis of pneumonia made? | No |
| | | Was an antibiotic started for treatment of pneumonia? | No |
| | | Concomitant antibiotic medication # | N/A |
| | XXXXXX | Was a chest assessment performed?/Reason if not assessed | Yes |
| | | Date/Time/Day performed | YYYY-MM-DD/HH:MM/## |
| | | Does chest x-ray show new or progressive infiltrates suggestive of pneumonia? | No |
| | | Has the subject been hospitalized for > 48 hours? | Yes |
| | | Has the subject received mechanical ventilation via an | |
| | | endotracheal or nasotracheal tube for >= 48 hours? | Yes |

Placebo

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

# Listing 16.2.6.9 Clinical Signs and Symptoms and Pneumonia Progression Pilot Rx Arm Amendment Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day<br>of Assessment/<br>Reason Not Done | Cough?/Rales?/<br>Percussion<br>Dullness? | Bronchial<br>Sounds?/<br>Egophony? | Suctioning?/<br>Ventilator? | Fever (>=38 C) | Purulent<br>Secretions | Dyspnea?/<br>Tachypnea | Hypoxemia?/<br>Supplemental O2 |
|---|---|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | xxxxx | YYYY-MM-DD/HH:MM/<br>## | Yes/Yes/<br>Yes | Yes/<br>No | Yes/<br>Yes | Yes | No | Yes/<br>No | Yes/<br>Yes |
| | XXXXXX | YYYY-MM-DD/HH:MM/<br>## | Yes/Yes/<br>Yes | Yes/<br>No | Yes/<br>Yes | Yes | No | Yes/<br>No | Yes/<br>Yes |

XXXXXX No/XXXXXXXXX

Placebo

Program Name: XXXX.sas Protocol Number: ASN100-201 Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM


Listing 16.2.6.10 Investigator Clinical Outcome of Pneumonia Pilot Rx Arm Amendment Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day<br>of Assessment/<br>Reason Not Done | Pneumonia Status | Continued Antibiotic<br>Therapy Required? | Antibiotic Therapy<br>Changed?* |
|---|---|---|---|---|---|
| ASN100 | | | | | |
| ###-##-## | XXXXXX | YYYY-MM-DD/HH:MM/## | Continues | Yes | |
| | XXXXXX | YYYY-MM-DD/HH:MM/## | Continues | Yes | |
| | Day 3 | YYYY-MM-DD/HH:MM/## | Continues | Yes | Yes |
| | XXXXXX | YYYY-MM-DD/HH:MM/## | Resolved | No | |
| | XXXXXX | YYYY-MM-DD/HH:MM/## | | | |
| ###-###-### | XXXXXX | YYYY-MM-DD/HH:MM/## | Continues | Yes | |
| | XXXXXX | YYYY-MM-DD/HH:MM/## | XXXXXXXXXXXXX | | |
| Placebo | | | | | |

Day = Study day and is based on first dose of study drug which is Day 1.  $\star$  Was antibiotic therapy changed within the first 48 hours based on insufficient therapeutic effect?

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.6.11 Hospitalization Course and Discharge Intent-to-Treat Population

| Treatment<br>Subject | Date/Time/Day<br>of Admission | Type of<br>Admission | ICU<br>Specify [1] | Discharged? | Date/Time/Day<br>of Discharge | Type of<br>Discharge |
|---|---|---|---|---|---|---|
| ASN100<br>###-###-### | YYYY-MM-DD/HH:MM/##<br>YYYY-MM-DD/HH:MM/## | ICU<br>Non-ICU | xxxxxxx | Yes<br>No | YYYY-MM-DD/HH:MM/## | xxxxxxxxxxxxxxxxx |
| ###-###-### | YYYY-MM-DD/HH:MM/## | ICU | Other: XXX | Yes | YYYY-MM-DD/HH:MM/## | Other: XXXXXXXXXXXXXXX |
| Placebo | | | | | | |

<sup>[1]</sup> MIC = Medical ICU, SICU = Surgical ICU, TICU = Trauma ICU, NICU = Neuro ICU, CCU = Coronary Care Unit, Other.

Protocol Number: ASN100-201


Program Name: XXXX.sas
Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.6.12 Anti-Drug Antibodies Sample Collection Intent-to-Treat Population

| Treatment<br>Subject | Visit | Collected? | Reason Sample Not Collected |
|----------------------|--------|------------|-----------------------------|
| ASN100 | | | |
| ###-##-### | Day 1 | Yes | |
| | Day 22 | No | Other: XXXXXX |
| | Day 90 | Yes | |
| ###-###-## | XXXXX | No | xxxxxxxxxxxx |
| Placebo | | | |

Protocol Number: ASN100-201


Program Name: XXXX.sas Run Date: MM/DD/YYYY HH:MM Data Last Modified: MM/DD/YYYY HH:MM

### Listing 16.2.6.13 Survival Status Intent-to-Treat Population

| ASN100 | |
|--------------------------------------------------|-------|
| ###-###-### Day ## YYYY-MM-DD/## Alive | |
| ###-###- Day ## YYYY-MM-DD/## Alive | |
| ###-###- Day ## Dead YYYY-MM-DD/## | |
| ###-### Day ## Unknown XXXXXXXXXXXXXXXXXXXXXXXXX | XXXX. |

Protocol Number: ASN100-201


Listing 16.2.7.1 Adverse Events

Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

Intent-to-Treat Population

| Treatment<br>Subject | VT: Verbatim Term<br>PT: Preferred Term<br>SOC:System Organ Class | Start Date/Time/Day<br>Stop Date/Time/Day<br>Duration (days) | SAE?/<br>TEAE?/<br>Severity | Related to<br>Study Drug | Action Taken/<br>Other Action Taken/<br>Outcome |
|---|---|---|---|---|---|
| ASN100 | | | | | |
| ###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/##/<br>## | No/<br>Yes/<br>SEVERE | NOT RELATED | XXXXXX/<br>XXXXXXXX/<br>FATAL |
| ###-###-### | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##/ | No/<br>No/<br>MILD | RELATED | XXXXXXXX/<br>XX /<br>NOT RECOVERED/NOT RESOLVED |
| | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD/HH:MM/##/<br>YYYY-MM-DD/HH:MM/##/<br>## | No/<br>Yes/<br>MODERATE | NOT RELATED | XXXXXXXX/<br>XXX<br>RECOVERED/RESOLVED WITH SEQUALE |

Placebo


Day = Study day and is based on the first dose of study drug which is day 1.

Duration is calculated using stop date of adverse event - start date of adverse event + 1.

A treatment-emergent adverse event (TEAE) is defined as an AE with a start date and time on or after the initiation of study drug administration. If the start time of an AE is missing, it is considered treatment emergent if it starts on the same date as the initiation

of study drug administration.

Protocol Number: ASN100-201


Listing 16.2.7.2 Serious Adverse Events

Intent-to-Treat Population

Program Name: XXXX.sas

Run Date: MM/DD/YYYY HH:MM

Data Last Modified: MM/DD/YYYY HH:MM

| Treatment<br>Subject | AE<br>Num | VT: Verbatim Term<br>PT: Preferred Term<br>SOC:System Organ Class | Birth Defect/<br>Significant<br>Disability | Death/<br>Autopsy/<br>Date/Day of Death | Hospitalization/<br>Life Threatening/<br>Other Medically<br>Important Event | Other<br>Possible<br>Causes | Event<br>Description |
|---|---|---|---|---|---|---|---|
| ASN100<br>###-###-## | # # | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No/<br>No | No/<br>No/<br>YYYY-MM-DD/## | No<br>Yes/<br>Yes | xxxxxxxxxxx | xxxxxxxxxxxxxxx |
| xxxxxxxxxx | #<br>XXXXX | VT: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No/ | No | Yes/<br>No/<br>Yes | xxxxxxxxxxxx | |
| Placebo | | | | | | | |


Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.8.1 Central Laboratory Parameters - Chemistry Intent-to-Treat Population

| Parameter (Unit) | Normal Range | Visit | Date/Time/Day<br>Collection | Result | Reference<br>Range [1] | Comments |
|---|---|---|---|---|---|---|
| XXXXXXX (XX) | ## - ### | XXXXX | YYYY-MM-DD/HH:MM/## | ### | LN | |
| | | XXXXX | YYYY-MM-DD/HH:MM/## | ### | LN | |
| | | XXXXX | YYYY-MM-DD/HH:MM/## | ### | N | |
| XXXXXXX (XX) | ## - ### | XXXXX | YYYY-MM-DD/HH:MM/## | ### | N | |
| | | XXXXX | YYYY-MM-DD/HH:MM/## | ### | N | |
| | | XXXXX | YYYY-MM-DD/HH:MM/## | ### | | |
| | XXXXXXX (XX) | XXXXXXX (XX) ## - ### | XXXXXXX (XX) ## - ### XXXXX<br>XXXXX<br>XXXXXX (XX) ## - ### XXXXX<br>XXXXXX | Parameter (Unit) Normal Range Visit Collection XXXXXXXX (XX) ## - ### XXXXX YYYY-MM-DD/HH:MM/## XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Parameter (Unit) Normal Range Visit Collection Result XXXXXXXX (XX) ## - ### XXXXXX YYYY-MM-DD/HH:MM/## #### XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Parameter (Unit) Normal Range Visit Collection Result Range [1] XXXXXXXX (XX) ## - ### XXXXX YYYY-MM-DD/HH:MM/## ## ## LN XXXXXX YYYY-MM-DD/HH:MM/## ## ## N XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

###-###-##

#### Placebo

<sup>[1]</sup> LN = Low Normal, LP = Low Panic, N = Normal, HN = High Normal, HP = High Panic, AB = Abnormal, SC = See Comment.

### The layouts of the following listings will be the same as listing 16.2.8.1:

Listing 16.2.8.2
Central Laboratory Parameters - Hematology
Intent-to-Treat Population

Listing 16.2.8.3
Central Laboratory Parameters - Urinalysis
Intent-to-Treat Population

Listing 16.2.8.4

Central Laboratory Parameters - Coagulation
Intent-to-Treat Population

Listing 16.2.8.5
Central Laboratory Parameters - Procalcitonin
Intent-to-Treat Population

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.8.6 Urine Pregnancy Test from Local Laboratory Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day of Urine Sample/<br>Reason Not Done | Result |
|---|---|---|---|
| ASN100<br>###-###-###<br>###-###-###<br>###-###-###<br>###-###-### | XXXXX<br>XXXXX<br>XXXXX | Other: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Negative<br>Negative |

#### Placebo

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.8.7 Vital Signs Intent-to-Treat Population

| Treatment<br>Patient | Visit | Date/Time/Day<br>of Collection/<br>Reason Not Done | Height<br>(cm) | Weight<br>(kg) | SBP<br>(mmHg) | DBP<br>(mmHg) | Pulse<br>(bpm) | Respiratory<br>Rate<br>(breaths/min) | Temp<br>(C)/<br>Time | рН | PaO2<br>(mmHg) | PaCO2<br>(mmHg) | SpO2<br>(%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ASN100 | | | | | | | | | | | | | |
| ###-###-### | SCR | YYYY-MM-DD/HH:MM/## | ## | ## | ### | ### | ## | ### | ##/HH:MM | ## | ### | ### | ## |
| | XXXXX | YYYY-MM-DD/HH:MM/## | | | ### | ### | ## | ### | ##/HH:MM | | | | ## |
| | XXXXX | YYYY-MM-DD/HH:MM/## | | | ### | ### | ## | ### | ##/HH:MM | ## | ### | ### | |
| | XXXXX | YYYY-MM-DD/HH:MM/## | | | ### | ### | ## | ### | ##/HH:MM | ## | ### | ### | |
| ###-###-### | SCR<br>XXXXX<br>XXXXX | Site Error<br>Other: XXXXXXXXXXXXXX<br>YYYY-MM-DD/HH:MM/## | | | ### | ### | ## | ### | ##/HH:MM | ## | ### | ### | ## |

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

#### Listing 16.2.8.8 12-Lead Electrocardiogram Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day<br>of Measurement/<br>Reason Not Done | HR | PR | QRS | QT | RR | Overall<br>Interpretation | Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|
| ASN100 | | | | | | | | | |
| ###-###-## | Screening | YYYY-MM-DD/HH:MM/## | ### | ### | ### | ### | ### | Abnormal | No |
| | Day 1 | YYYY-MM-DD/HH:MM/## | ### | ### | ### | ### | ### | Normal | |
| | Day ## | Other: XXXX | | | | | | | |
| | Day ## | Subject Refused | | | | | | | |
| ###-###-## | Screening | Site Error | | | | | | | |
| | Day 1 | YYYY-MM-DD/HH:MM/## | ### | ### | ### | ### | ### | Normal | |
| | Day ## | YYYY-MM-DD/HH:MM/## | ### | ### | ### | ### | ### | Normal | |
| | Day ## | YYYY-MM-DD/HH:MM/## | ### | ### | ### | ### | ### | Not Evaluable | |

#### Placebo

 $\mbox{\tt Day} = \mbox{\tt Study} \mbox{\tt day} \mbox{\tt and}$  is based on first dose of study drug which is  $\mbox{\tt Day}$  1. Note: Unit of HR is bpm, and units of other measurements are msec.

143

Protocol Number: ASN100-201


Run Date: MM/DD/YYYY HH:MM
Data Last Modified: MM/DD/YYYY HH:MM

Program Name: XXXX.sas

### Listing 16.2.8.9 Physical Examination Intent-to-Treat Population

| Treatment<br>Subject | Visit | Date/Time/Day<br>Performed/<br>Reason Not Done | Overall<br>Assessment* | Specify<br>Abnormalities |
|---|---|---|---|---|
| ASN100 | | | | |
| ###-##-## | Screening | YYYY-MM-DD/HH:MM/## | Normal | |
| | Day 1 | YYYY-MM-DD/HH:MM/## | Abnormal and CS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Day ## | YYYY-MM-DD/HH:MM/## | Abnormal but NCS | |
| | XXXXXX | Other: XXXXXXX | | |
| ###-##-## | Screening | Site Error | | |
| | Day 1 | YYYY-MM-DD/HH:MM/## | Abnormal and CS | XXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXX | Subject Refused | | |
| lacebo | | | | |

Day = Study day and is based on first dose of study drug which is Day 1.

<sup>\*</sup> CS = Clinically Significant, NCS = Not Clinically Significant.